## The GlaxoSmithKline group of companies

 Division
 : Worldwide Development

 Information Type
 : Reporting and Analysis Plan

Title : Reporting and Analysis Plan for 201749: A 24-week treatment, multi-center, randomized, double-blind, double-dummy, parallel group study to compare Umeclidinium/Vilanterol, Umeclidinium, and Salmeterol in subjects with chronic obstructive pulmonary disease (COPD)

Compound Number : GSK2592356 (GSK573719+GW642444)

Effective Date : 18-JUL-2018

## **Description:**

• The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the main Clinical Study Report for Protocol 201749.

## **RAP Author(s):**

## Author

PPD

Principal Statistician, RD PCPS Qsci Clinical Statistics

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|-----------------------------------|-------------|-----------------|
| PPD | 05-JUL-2018 | Esig |
| Clinical Development Director | 03-JUL-2018 | Esig |
| PPD | 17-JUL-2018 | Esig |
| Operational Study Lead | 17-JUL-2018 | Esig |
| PPD | 18-JUL-2018 | Esig |
| Manager, Clinical Data Management | 10-JUL-2016 | Esig |
| PPD | 05-JUL-2018 | Email |
| GMAL | 03-JUL-2018 | Ellian |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Senior Statistics Director, RD PCPS Qsci Clinical Statistics | 05-JUL-2018 | Esig |
| PPD Programming Manager, RD PCPS Qsci Clinical Statistics | 13-JUL-2018 | Esig |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 6 |
| 2. | STIM | MARY OF KEY PROTOCOL INFORMATION | Q |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objectives and Endpoints | ٥٥ |
| | 2.2. | Study Objectives and Endpoints | |
| | 2.3.<br>2.4. | Statistical Hypotheses | |
| | 2.4. | Statistical hypotheses | 13 |
| 3. | DI AN | INED ANALYSES | 1/ |
| J. | 3.1. | Final Analyses | |
| | J. I. | Filial Allalyses | 14 |
| 4. | ANAL | YSIS POPULATIONS | 14 |
| | 4.1. | Protocol Deviations | 15 |
| 5. | CON | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates and Other Strata | |
| | | 5.4.1. Covariates and Other Strata | 17 |
| | 5.5. | Multiple Comparisons and Multiplicity | 17 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 17 |
| _ | 07115 | NV DODUK ATION ANALYOFO | 40 |
| 6. | | DY POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | |
| | | 6.1.1. Disposition | |
| | | 6.1.2. Medical Conditions | |
| | | 6.1.3. Concomitant Medications | |
| | | 6.1.4. Screening Lung Function Tests | 19 |
| | | 6.1.5. GOLD Grade/Categories, Reversibility and long-acting | |
| | | bronchodilator usage Stratum | |
| | | 6.1.6. Maintenance Naive | 19 |
| 7. | PRIM | ARY STATISTICAL ANALYSES | 19 |
| • | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | |
| | | 7.1.5.1. Statistical Methodology Specification | |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | Chatogy for interestrictit (1 oot i tarradinization) Events | |

| | | 7.2.5. | Statistical Analyses / Methods | |
|---|---|---|---|---|
| | 7.3. | Evnlorat | 7.2.5.1. Statistical Methodology Specification | |
| | 1.5. | 7.3.1. | Endpoint / Variables | |
| | | 7.3.1. | Summary Measure | |
| | | 7.3.3. | Population of Interest | |
| | | 7.3.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.3.5. | Statistical Analyses / Methods | |
| | | 7.0.0. | 7.3.5.1. Statistical Methodology Specification | |
| | 7.4. | Subgrou | ip Analyses | |
| 8. | | | YSES | |
| | 8.1. | | Events Analyses | |
| | 8.2. | | Events of Special Interest Analyses | |
| | 8.3. | Clinical I | Laboratory Analyses | 35 |
| 9. | REFE | RENCES | | 36 |
| ٥. | IXLIL | INLINOLO | | |
| 10. | APPE | NDICES. | | 37 |
| | 10.1. | | x 1: Schedule of Activities | |
| | | | Protocol Defined Schedule of Events | |
| | 10.2. | | x 2: Assessment Windows | |
| | | | Definitions of Assessment Windows for Analyses | |
| | 10.3. | | x 3: Study Phases and Treatment Emergent Adverse | 41 |
| | | 10.3.1. | | |
| | | 10.3.2. | Study Phases for Adverse Events and All Other Data | |
| | | | Recorded in Logs (excluding Concomitant Medications) | 42 |
| | | 10.3.3. | Treatment Emergent Flag for Adverse Events and | |
| | | | Exacerbations | 42 |
| | 10.4. | Appendi | ix 4: Data Display Standards & Handling Conventions | 43 |
| | | 10.4.1. | Reporting Process | |
| | | 10.4.2. | Reporting Standards | 43 |
| | 10.5. | Appendi | x 5: Derived and Transformed Data | 45 |
| | | 10.5.1. | General | |
| | | 10.5.2. | Study Population | 45 |
| | | 10.5.3. | Efficacy | |
| | | 10.5.4. | Safety | |
| | 10.6. | Appendi | x 6: Reporting Standards for Missing Data | 60 |
| | | 10.6.1. | | |
| | | 10.6.2. | | |
| | | | 10.6.2.1. Handling of Missing Dates | |
| | | | 10.6.2.2. Handling of Partial Dates | 61 |
| | | | 10.6.2.3. Handling of Missing Data for Statistical | 0.4 |
| | 40 = | | Analysis | 61 |
| | 10.7. | | x 7: Abbreviations & Trade Marks | |
| | | 10.7.1. | Abbreviations | |
| | 40.0 | 10.7.2. | Trademarks | |
| | 10.8. | | ix 8: List of Data Displays | |
| | | 10.8.1. | Data Display Numbering Deliverables | |
| | | | Study Population Tables | |

# 2018N377698\_00 201749

## CONFIDENTIAL

| 10.8.4. | Efficacy Tables | 67 |
|----------|-------------------------|----|
| | Efficacy Figures | |
| | Safety Tables | |
| | Safety Figures | |
| 10.8.8. | ICH Listings | 78 |
| 10.8.9. | Non-ICH Listings | 84 |
| 10.8.10. | Maintenance Naive | 84 |
| 10.8.1. | Study Population Tables | 84 |
| 10.8.2. | Efficacy Tables | 86 |
| 10.8.3. | Efficacy Figures | 91 |
| | Safety Tables | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|------------------------------------|-------------|-----------------|
| GlaxoSmithKline Document<br>Number | Date | Version |
| 2016N277425_00 | 2016-SEP-13 | Original |
| 2016N277425_01 | 2017-FEB-07 | Amendment No. 1 |

This protocol amendment was created to make the following changes:

Regulatory Agency Identifying Number(s): A typographical error in the EudraCT no. corrected. IND no. added

Section 4.1 and Section 4.4: Typographical errors and inconsistencies corrected

Inconsistencies between Section 4.4, Section 7.3.1.5 and Section 7.1 revised

Section 7.1 Time and Events table:

Un-intentional deletion of the ("x") were added to confirm that concomitant medications should be reviewed at every clinic visit was corrected.

Increased the visit window

Typographical error and inconsistencies corrected as described in Appendix 9, Section 12.9.

Section 7.2.2 Critical procedures performed at Screening (Visit 1): To clarify that height and weight are collected at V1 "Height and weight" added

Section 7.3.2 Spirometry: "At Screening, before the morning dose of usual COPD medication(s)" added.

Section 7.3.7: Physical activity monitor (study subset) Inconsistency between Section 1, Section 4.1 and Section 7.3.7 revised

| 2016N277425_02 | 2017-FEB-21 | Amendment No. 2 Canada |
|----------------|-------------|------------------------|
| | | ONLY |

This protocol amendment was created to comply with Health Canada guidelines. They require pharmaceutical manufacturers to expeditiously report domestic cases of unusual failure in efficacy (UFIE) for new drugs to the Marketed Health Products Directorate (MHPD) within 15 days of first notification.

Changes were made to Section 7.4.1 and Appendix 4.

| Revision Chronology: | | |
|------------------------------------|-------------|-----------------|
| GlaxoSmithKline Document<br>Number | Date | Version |
| 2016N277425_03 | 2017-APR-18 | Amendment No. 3 |

This protocol amendment was created to make the following changes:

- Clarifications concerning study design, stratification, permitted and prohibited COPD medications, stopping criteria, visit windows, chest x-rays performed in the context of the protocol and site professional expertise
- Rate of COPD exacerbations from tertiary endpoints to exploratory endpoints
- Addition of an inclusion criterion specific to France
- Integration of Canadian Amendment 2
- Correction of typographical errors and inconsistencies

Note there is a separate RAP to cover the required analyses for the German Federal Joint Committee (G-BA).

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | <ul> <li>An additional population<br/>has been defined, the<br/>Activity Monitoring (AM)<br/>Population, which will<br/>comprise all subjects in<br/>the ITT population who<br/>provide data from at least<br/>one activity monitoring<br/>session.</li> </ul> | Population needed for<br>subset of subjects<br>participating in Activity<br>Monitoring. |
| | All other Endpoints promoted to secondary endpoints | Study aims have<br>developed since protocol<br>and thus previous<br>endpoints classed as<br>'other' have further<br>importance |
| | An analysis by Maintenance Naive (MN) and Non-Maintenance Naive subgroups have been included. | To investigate prospectively the 1st line use of LAMA/LABA in all symptomatic subjects (no existing data I the literature to our knowledge) |
| | <ul> <li>An analysis of ratio of<br/>trough FEV1 to baseline<br/>trough FEV1</li> </ul> | To investigate trough FEV1 ratio change from baseline |
| Intent-to-treat ICS free (ITT ICS free) | Population excluded. | G-BA analysis to be conducted on the ITT population due to a change in G-BA guidance. |
| To compare albuterol/salbutamol use captured in the eDiary with the electronic metered dose inhaler (eMDI) Device as data allow | Not included in this RAP. | Will be included in a supplementary RAP if deemed necessary. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| To compare physical activity levels, ER-S, rescue medication use, hospital exacerbations and mortality in subjects with and without a CID | To compare ER-S,<br>rescue medication use,<br>hospital exacerbations<br>and mortality in subjects<br>with and without a CID | Physical activity levels<br>will not be assessed via<br>CID due to a smaller<br>subset of subjects. |

There were changes to the originally planned populations specified in the protocol (Dated: 13-SEP-2016) and Table 1.

# 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | Primary |
| To compare the effect of UMEC/VI<br>(62.5/25 mcg once daily) with UMEC<br>(62.5 mcg once daily) on lung function | Change from baseline in trough Forced Expiratory Volume in One Second (FEV <sub>1</sub> ) at week 24 |
| Secondary | Secondary |
| To compare UMEC/VI (62.5/25 mcg once daily), UMEC (62.5 mcg once daily) with salmeterol (50 mcg twice daily) on patient reported outcomes | Change from baseline in self administered computerised (SAC) transient dyspnea index (TDI) |
| (PROs) | <ul> <li>Percentage of TDI responders according to SAC<br/>TDI score. A responder is defined as a ≥1 unit<br/>improvement in SAC TDI score</li> </ul> |
| | Assessment of respiratory daily symptoms over<br>24 weeks using Evaluating Respiratory<br>Symptoms- COPD (E-RS) and its subscales<br>(breathlessness, cough and sputum and chest<br>symptoms) |
| | <ul> <li>Percentage of E-RS responders according to E-RS score (defined as reduction in E-RS score of ≥2 or ≥3.35 units) from baseline</li> </ul> |
| | Change from baseline in St George's Respiratory<br>Questionnaire (SGRQ-C) |
| | Percentage of responders according to SGRQ-C total score (defined as a 4 point or greater reduction from baseline) |
| | Change from baseline in COPD assessment test (CAT) |
| | Percentage of responders according to CAT |

| Objectives | Endpoints |
|---|---|
| | (defined as a ≥2 unit improvement in score from baseline) |
| To compare UMEC/VI (62.5/25 mcg once daily), UMEC (62.5 mcg once daily) with salmeterol (50 mcg twice daily) on other COPD efficacy measures To compare UMEC/VI (62.5/25 mcg once daily), UMEC (62.5 mcg once daily) with salmeterol (50 mcg twice daily) on other COPD efficacy measures | <ul> <li>Ratio to baseline of trough Forced Expiratory Volume in One Second (FEV1)</li> <li>Time to first mild, moderate or severe exacerbation</li> <li>Time to first moderate or severe exacerbation</li> <li>Time to first severe exacerbations</li> <li>Time to first clinically important deterioration (CID) composite endpoint</li> <li>Time to first clinically important deterioration composite endpoint excluding FEV1 (Exacerbation, SGRQ, TDI, CAT)</li> <li>Rescue albuterol/salbutamol use, (percentage of rescue-free days and mean number of Inhalations/day) captured by the electronic diary (eDiary) over 24 weeks</li> <li>Inspiratory capacity (IC)</li> <li>Forced Vital capacity (FVC)</li> <li>Change from baseline in trough FEV1</li> </ul> |
| | <ul> <li>Change from baseline in global impression of disease severity</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Safety | Safety |
| To evaluate safety and tolerability of<br>UMEC/VI (62.5/25 mcg once daily),<br>UMEC (62.5mcg once daily) and<br>salmeterol 50mcg twice daily) | Incidence of adverse events |
| Exploratory | Exploratory |
| To explore the effect of UMEC/VI (62.5/25 mcg once daily), UMEC (62.5 mcg once daily) with salmeterol (50 mcg twice daily) on rate of COPD exacerbation | <ul> <li>Rate of mild, moderate or severe exacerbations</li> <li>Rate of moderate or severe exacerbation</li> </ul> |
| To explore the effect of UMEC/VI (62.5/25 mcg once daily), UMEC (62.5 mcg once daily) with salmeterol (50 mcg twice daily) on physical activity | Change from baseline in physical activity |
| To investigate the CID composite<br>endpoint ability to predict short term<br>outcomes | <ul> <li>To compare ER-S, rescue medication use,<br/>hospital exacerbations and mortality in subjects<br/>with and without a CID</li> </ul> |

# 2.3. Study Design



# **Overview of Key Study Design Features**

## **Design Features:**

- Multi-centre, randomized, double blind, double dummy, 3-arm parallel group study to compare Umeclidinium/Vilanterol, Umeclidimium, and Salmeterol in subjects with chronic obstructive pulmonary disease (COPD).
- Approximately 3232 subjects will be screened, such that 2424 subjects will be randomized and approximately 2181 evaluable subjects complete the study.
- Eligible subjects will be stratified by country, long-acting bronchodilator usage during the run-in (none or one long-acting bronchodilator per day) and activity subset (activity subset or no activity subset), and randomized in a ratio of 1:1:1 to UMEC/VI inhalation powder (62.5/25 mcg once daily) administered via the ELLIPTA inhaler, or UMEC (62.5 mcg once daily) administered via the ELLIPTA or salmeterol (50 mcg BID) administered via the DISKUS. Note the activity subset was only included as a randomisation stratification group for logistical purposes.
- A subset of subjects up to 150 per treatment arm will undergo assessment of their physical activity measured through a physical activity monitor (Actigraph GT9X) worn for 7 days from Screening (Visit 1), for 7 days from Randomisation (Visit 2), 7 days from Visit 3, and for 7 days prior to last clinic Visit (Visit 5).
- The total duration of subject participation in the study will be approximately 29 to 35 weeks consisting of 6 weeks prescreening if necessary, 4 weeks run-in, 24 week treatment and one week Follow-Up.

#### Dosing:

- The following study medications will be used in this study:
  - UMEC/VI 62.5/ 25mcg administered via ELLIPTA
  - UMEC 62.5 mcg administered via ELLIPTA
  - Salmeterol 50 mcg administered via DISKUS
  - Placebo via ELLIPTA
  - Placebo via DISKUS

Subjects will be instructed to take one dose of medication each morning from the ELLIPTA (one inhalation equals one dose), and one dose in the morning and one in the evening from the DISKUS.

The ELLIPTA will provide a total of 30 doses and the DISKUS will provide a total of 60 doses.

| Overview of Key Study Design Features | |
|---|---|
| Treatment Assignment: | Subjects will be randomly assigned to one of the blinded stud<br>treatment regimens in equal proportion (ratio of 1:1:1): |
| | <ul> <li>UMEC/VI 62.5/25 mcg once daily via ELLIPTA + placebo<br/>twice daily via DISKUS</li> </ul> |
| | <ul> <li>UMEC 62.5 mcg once daily via ELLIPTA + placebo twice<br/>daily via DISKUS</li> </ul> |
| | <ul> <li>Salmeterol 50 mcg twice daily via DISKUS + placebo once daily via ELLIPTA</li> </ul> |
| | GSK RandAll NG used to generate randomisation schedules. |
| | • Centralised randomisation within country using GSK RAMOS NG for treatment allocation. |
| | <ul> <li>Stratified by long-acting bronchodilator usage during run-in (none<br/>or one long-acting bronchodilator per day), country and<br/>activity subset (activity subset or no activity subset). Note the<br/>activity subset was only included as a randomisation stratification<br/>group for logistical purposes.</li> </ul> |
| Interim Analysis | No interim analysis will be performed. |

# 2.4. Statistical Hypotheses

The primary purpose of this study is to demonstrate improvements in lung function for subjects treated with UMEC/VI compared with UMEC for 24 weeks.

The primary endpoint is change from baseline in trough FEV<sub>1</sub> at Week 24. The null hypothesis is no difference between treatment groups (H0:  $\mu$ T –  $\mu$ S = 0), with the alternative hypothesis that there is a difference between treatment groups (H1:  $\mu$ T –  $\mu$ S  $\neq$  0), where  $\mu$ T is the mean change from baseline for UMEC/VI and  $\mu$ S is the mean change from baseline for UMEC.

In order to account for multiplicity across treatment comparisons and endpoints, a step-down closed testing procedure will be applied whereby inference for secondary endpoints or treatment comparisons are dependent upon statistical significance having been achieved for the primary comparison. If the primary comparison is significant i.e. the associated p-value for UMEC/VI versus UMEC for change from baseline in trough FEV1 at Week 24 is below 0.05, this will allow inference of treatment comparisons (UMEC/VI versus UMEC on all secondary endpoints, and UMEC/VI versus Salmeterol and UMEC versus Salmeterol on all primary and secondary endpoints), which will be declared statistically significant if the associated p-value is below 0.05.

## 3. PLANNED ANALYSES

## 3.1. Final Analyses

The final planned analyses of the study will be performed after the completion of the following sequential steps (for this Clinical Data Interchange Standards Consortium [CDISC] study):

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final System Independent (SI) database release has been declared by Data Management (DM).
- 3. SI data to SDTM data conversion has completed by Conversion Service and quality control of unblinded SDTM has completed by DM.
- 4. All criteria for unblinding the randomization codes have been met.
- 5. Randomization codes have been distributed according to [RandAll NG].
- 6. Database freeze on SDTM datasets has been declared by DM

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All<br>Subjects<br>Enrolled<br>(ASE) | All subjects for whom a record exists in the study database, including screen failures and any subject who was not screened but experienced an SAE between the date of informed consent and the planned date of the Screening visit. | <ul> <li>Subject Disposition</li> <li>Reasons for<br/>withdrawal prior to<br/>randomisation</li> <li>Inclusion, exclusion<br/>and randomisation<br/>criteria deviations</li> <li>SAEs for non-<br/>randomised subjects</li> </ul> |
| Intent-to-<br>treat (ITT) | <ul> <li>All randomized subjects (excluding those who were randomized in error) who received at least one dose of study medication. A subject who is recorded as a screen or run-in failure and also randomized will be considered to be randomized in error. Any other subject who receives a randomization number will be considered to have been randomized.</li> <li>Displays will be based on the treatment to which the subject was randomized</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li><li>Safety</li></ul> |
| Activity<br>Monitoring<br>(AM) | <ul> <li>All subjects in the ITT population who provide data from at least one activity monitoring session.</li> <li>Displays will be based on the treatment to which the subject was randomized</li> </ul> | Activity Monitoring |

#### 1. NOTE:

 Please refer to Section 10.8 Appendix 8: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Protocol deviations (PDs) will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP).
- Data will be reviewed by SDL prior to SDTM DBF to ensure all important deviations are captured and categorized on the protocol deviations dataset (except for the PD of taking incorrect treatment).
- Subjects who received an incorrect container will be captured as an important protocol deviation. Whether or not the incorrect container contains incorrect treatment will be identified following DBF in the Analysis Data Model (ADaM) dataset.
- Important protocol deviations (as identified in the PDMP) will be summarized and listed.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporting | |
| Code | Description | Description | Order in TFL |
| 1 | UMEC/VI 62.5/25 mcg once daily via ELLIPTA + placebo twice daily via DISKUS | UMEC/VI 62.5/25 | 1 |
| 2 | UMEC 62.5 mcg once daily via<br>ELLIPTA + placebo twice daily via<br>DISKUS | UMEC 62.5 | 2 |
| 3 | Salmeterol 50 mcg twice daily via DISKUS + placebo once daily via ELLIPTA | SAL 50 | 3 |

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest predose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Endpoint | Baseline derivation |
|---|---|
| Trough FEV <sub>1</sub> , FVC and IC | The mean of the values measured at 30 min and 5 min predose on Day 1. If the actual time of an assessment is after the time of dosing on Day 1, the value at that assessment will be |

| Endpoint | Baseline derivation |
|---|---|
| | set to missing prior to calculating baseline. |
| | If one of the values is missing then the baseline will be the single remaining value; otherwise the baseline will be the mean of the two values. |
| TDI | BDI assessment taken prior to dosing on Day 1. |
| | The baseline dyspnea index (BDI) focal score will be calculated as the sum of the ratings recorded for each of the three individual scales (Functional Impairment, Magnitude of Task, Magnitude of Effort). Each of these scales has five possible scores ranging from 0 to 4 (with lower scores indicating more impairment), so the range of the BDI focal score is 0 to 12. If a score is missing (or has a value of W, X or Y) for any of the three scales, then the BDI focal score will be set to missing. |
| E-RS and subscale scores | Average of measurements from day -28 to day -1 inclusive; at least 16 days must be non-missing. |
| Physical activity | Average of measurements prior to randomisation; at least 3 days must be non-missing. |
| Rescue Use - Mean Number of<br>Puffs of Rescue Medication<br>Per Day and Percentage of<br>Rescue-free Days Over Weeks<br>1-24 captured using e-diary | The total puffs of rescue for each day will be calculated as number of salbutamol puffs. If the number of puffs is missing then the total puffs will be set to missing for that day. The baseline number of inhalations is calculated using the mean number of total inhalations and the baseline percentage rescue use is calculated from the percentage of rescue free days as the average of measurements from day -28 to day -1 inclusive; at least 14 days must be non-missing. |
| Rescue Use - Mean Number of<br>Occurrences of Rescue<br>Medication Per Day and | The total occurrences, defined as =>1 puff within a 2 minute time window, of rescue for each day will be calculated. |
| Percentage of Rescue-free Days Over Weeks 1-24 captured using e-MDI | The baseline is calculated using the mean number of occurrences and the baseline percentage rescue use is calculated from the percentage of rescue free days as the average of measurements from the first date of sensor sync to the last date of sensor sync (per sensor subject combination) up until the day prior to first dose. |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

- This study will be randomized centrally within country.
- It is likely that many centres will enrol a very small number of subjects and so rather than
  adjusting for centre in the statistical analyses, a geographical region will be used. This will
  consist of all centres within a similar geographical region.
- Country is determined by the location of the centre, as entered into GSK systems by the site monitor. The CENTREID variable will be used to identify and group centres.
- Geographical Region will be used wherever geographical region is included and defined as follows:

| South America | North America | EU | Other |
|---------------|---------------|-------------|--------------|
| Argentina | Canada | France | Australia |
| Mexico | US | Germany | South Africa |
| | | Italy | |
| | | Netherlands | |
| | | Spain | |
| | | Sweden | |

#### 5.4. Examination of Covariates and Other Strata

## 5.4.1. Covariates and Other Strata

- Randomization is stratified by long-acting bronchodilator usage during the run-in (none
  or one long-acting bronchodilator per day) and long-acting bronchodilator usage will be
  included as a covariate in all statistical models. The no. of bronchodilators per day during
  run-in be re-derived and used for analysis. The randomized stratum from RAMOS and
  reported on the eCRF will be listed only.
- Other covariates will be included for specific analyses as detailed in model specifications in Section 7 and Section 8.

# 5.5. Multiple Comparisons and Multiplicity

See Section 2.4 for details on inferences that can be drawn on primary, secondary and 'other' endpoints.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.2 | Appendix 2: Assessment Windows |
| 10.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Reporting Standards for Missing Data |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the ITT population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 8: List of Data Displays

## 6.1.1. Disposition

The study population summary will show the number of subjects overall who were enrolled, the number of pre-screen failures, the number of screen failures and the number with each reason for screen failure, the number of run-in failures each reason the number with each reason for run-in failure and the number of subjects in each treatment group and overall who were randomized, in the ITT population. Of those in the ITT population the number and percentage of subjects in the AM population will be presented by treatment and overall.

The end of study record summary shows the number of subjects who completed the study as well as the number who withdrew early from the study along with reasons for early withdrawal.

The summary of study treatment status shows the number of subjects who completed study treatment as well as the number who stopped study treatment prior to the end of the study, along with the reasons for discontinuation.

#### 6.1.2. Medical Conditions

The number and percentage of subjects reporting each current medical condition will be presented by randomized treatment group and overall. All medical conditions must be summarised on this table regardless of frequency.

This will be repeated for past medical conditions.

#### 6.1.3. Concomitant Medications

Medications that have been stopped prior to Screening will be listed and not be included in any summary tables.

Medications not taken for an exacerbation will be summarised by Anatomical-Therapeutic-Chemical (ATC) level 1 and ingredient. COPD medications given for an exacerbation will be summarised by Respiratory Medication Class (RMC).

Medications taken for an exacerbation and those not taken for an exacerbation will be listed separately. Both listings will indicate in which study phases each medication was taken (pre-treatment and/or on-treatment and/or post-treatment)

## 6.1.4. Screening Lung Function Tests

Pre- and post-salbutamol FEV<sub>1</sub>, FVC and FEV<sub>1</sub>/FVC ratio, post-salbutamol FEV<sub>1</sub> as a percentage of predicted normal and FEV<sub>1</sub> reversibility to salbutamol (expressed in mL and as a percentage) at Screening will be summarised by treatment group and overall.

# 6.1.5. GOLD Grade/Categories, Reversibility and long-acting bronchodilator usage Stratum

The number and percentage of subjects in each GOLD Grade 1-4 and GOLD Category A-D using CAT, the number and percentage of subjects classified as Reversible/Non-reversible to salbutamol at Screening and the number and percentage of subjects in each stratum (none or one long-acting bronchodilators per day) based on the long-acting bronchodilator usage during run-in (all defined in Section 10.5.2) will be presented by treatment group and overall.

#### 6.1.6. Maintenance Naive

Summary Maintenance Naive and Non-Maintenance Naive status will be presented by treatment group and overall.

#### 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoint / Variables

Trough FEV<sub>1</sub> at Week 24

## 7.1.2. Summary Measure

Mean change from baseline

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the ITT population,.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

An intercurrent event considered to have an impact on the estimand for the ITT population analysis is:

• Discontinuation of randomised treatment

• The primary treatment effect to be estimated for the ITT population will be the hypothetical effect if all subjects had stayed on their randomised treatment.

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.1.5.1. Statistical Methodology Specification

#### **Primary Statistical Analysis**

## **Endpoint**

• Change from Baseline in trough FEV<sub>1</sub> at Week 24 (results for trough FEV<sub>1</sub> at all other time points and other treatment comparisons will be obtained from the same analysis even though those are not the primary endpoint)

## **Model Specification**

- Trough FEV<sub>1</sub> at Week 24 will be analysed for the ITT population using a mixed model repeated measures (MMRM) including data recorded at each of Week 4, Week 12 and Week 24.
- The following covariates will be included in the model: baseline FEV<sub>1</sub>, geographical region, stratum (no. of bronchodilators per day during run-in), visit, treatment, visit by baseline and visit by treatment interactions, where visit is nominal.
- Two models will be fitted; one with a response variable of trough FEV<sub>1</sub>, and one with a response variable of change from baseline in trough FEV<sub>1</sub>.
- While missing data are not explicitly imputed in the primary MMRM analyses, there is an underlying assumption that the data are missing at random.
- The Kenward and Roger method (KR) for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- In the event the model fails to run using the KR method, then the residual method will be used instead.
- An unstructured covariance structure for the R matrix will be used by specifying 'type='UN' on the REPEATED line.
- Results for all time points where data are scheduled to be collected and all treatment comparisons will be included in the analysis and presented in the displays.

## **Model Checking & Diagnostics**

 Model assumptions will be applied but appropriate adjustments may be made based on the data.

## **Primary Statistical Analysis**

- Normality assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriately transformed data.

#### **Model Results Presentation**

- Least squares (LS) mean and LS mean changes from baseline with their corresponding standard errors (SEs) will be presented for each treatment by visit, together with estimated treatment differences (UMEC/VI 62.5/25 vs. UMEC 62.5, UMEC/VI 62.5/25 vs Salmeterol and UMEC 62.5 vs Salmeterol), corresponding 95% CIs and p-values.
- A plot of LS mean changes from baseline and 95% CIs for each treatment by visit will be generated.
- A plot of LS mean treatment differences and 95% CIs between the treatment groups by visit will also be generated.
- The type III tests of fixed effects and the covariance parameter estimates from the model will be presented in two tables.

## **Summary Results Presentation**

- Summary of baseline FEV<sub>1</sub> will be presented by treatment for all subjects.
- A box plot and an empirical distribution function plot of change from baseline in trough FEV<sub>1</sub> at Week 24 will be produced.
- Summary statistics for raw and change from baseline in trough FEV<sub>1</sub> at each visit and for each treatment will be presented on the same table.

## **Sensitivity and Support Statistical Analysis**

- An assessment of whether the effect of treatment is modified by the interaction with o Baseline FEV<sub>1</sub>
  - o Geographical Region
  - o Stratum (no. of bronchodilators per day during run-in) will be made (for primary endpoint only for the ITT population only) by fitting separate MMRM models including an additional term for treatment by each covariate. The interaction term will be tested at the 10% significance level.
- For factors with two levels or continuous factors i.e. Baseline FEV<sub>1</sub> and Stratum, interactions with treatment will be investigated by fitting a model with the same terms as the main model, and adding in treatment by factor by Visit interaction. Contrast statements will be used to obtain the p-value for the treatment by factor interaction at Week 24. If that p-value is >=0.10 the interaction will be considered not significant. If the p-value is <0.10, further investigation will be performed, for example running analysis by each level of the factor, or for subgroups

- above and below the median.
- For factors with more than 2 levels i.e. Geographical Region, the overall interaction of factor by treatment will be investigated by fitting a model with the same terms as the main model, and adding in treatment by factor interaction. The p-value for the overall treatment by factor interaction will be obtained. If that p-value is >=0.10 the interaction will be considered not significant. If the p-value is <0.10 then the analysis will be repeated including the treatment by factor by visit interaction and the p-value for the interaction on Week 24 obtained. If that p-value is >=0.10 the interaction will be considered not significant. If the p-value is <0.10 then the factor will be dichotomised for example US vs. non-US and EU vs. non-EU for geographical region interactions (several different dichotomies may be explored). A model will be fitted with the same terms as the main model, and adding in treatment by dichotomized factor by Visit interaction, and contrast statements will be used to obtain the p-value for the treatment by dichotomized factor interaction on Week 24. If that p-value is >=0.10 the interaction will be considered not significant. If the p-value is <0.10, further investigation will be performed, for example running analysis by each level of the factor.

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

- 1) SAC TDI focal score
- 2) Assessment of respiratory daily symptoms using E-RS and its subscales
- 3) Change from baseline in SGRQ
- 4) Change from baseline in CAT
- 5) Proportion of responders according to SAC TDI focal score
- 6) Proportion of responders according to E-RS total and subscale scores
- 7) Proportion of responders according to SGRQ total score
- 8) Proportion of responders according to CAT score
- 9) Time to first on-treatment mild/moderate/severe COPD exacerbation
- 10) Time to first on-treatment moderate/severe COPD exacerbation
- 11) Time to first on-treatment severe COPD exacerbation
- 12) Time to CID composite endpoint (including individual components)
- 13) Time to CID composite endpoint excluding FEV1 (including individual components)
- 14) Mean number of inhalations of rescue use per day (using eDiary)
- 15) Percentage of rescue-free days (using eDiary)
- 16) Trough FEV1 ratio to baseline
- 17) Trough FVC
- 18) Trough IC
- 19) Subject global rating of change in COPD severity

## 7.2.2. Summary Measure

- 1) Mean change from BDI score
- 2) Mean change from baseline
- 3) Mean change from baseline
- 4) Mean change from baseline
- 5) Odds ratio
- 6) Odds ratio
- 7) Odds ratio
- 8) Odds ratio
- 9) Hazard ratio
- 10) Hazard ratio
- 11) Hazard ratio
- 12) Hazard ratio
- 13) Hazard ratio
- 14) Mean change from baseline
- 15) Mean change from baseline
- 16) Ratio of trough FEV1 to baseline FEV1
- 17) Mean change from baseline
- 18) Mean change from baseline
- 19) Odds ratio

## 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the ITT population, unless otherwise specified.

## 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

All endpoints will use the same strategy for intercurrent events as defined in Section 7.1.4.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.2.5.1. Statistical Methodology Specification

#### TDI, E-RS, SGRQ-C and CAT Scores

## Secondary Statistical Analysis

#### **Endpoints**

- SAC TDI focal score
- Assessment of respiratory daily symptoms using E-RS and its subscales
- Change from baseline in SGRQ
- Change from baseline in CAT

## Model Specification, Checking and Results Presentation

- Similar to trough FEV1 in Section 7.1.5.1.
- For TDI one model will be fitted with a dependent variable of TDI and BDI in place of baseline.
- For E-RS and subscales, all 4-weekly mean scores will be included in the analysis.

## Responders according to TDI, E-RS, SGRQ-C and CAT Scores

#### **Secondary Statistical Analysis**

#### **Endpoints**

- Proportion of responders according to TDI focal score
- Proportion of responders according to E-RS total score
- Proportion of responders according to E-RS Breathlessness score
- Proportion of responders according to E-RS Cough & Sputum score
- Proportion of responders according to E-RS Chest Symptoms score
- Proportion of responders according to SGRQ total score
- Proportion of responders according to CAT score

#### **Model Specification**

- The proportion of responders will be analyzed using a generalized linear mixed model with treatment as an explanatory variable and visit, baseline score, stratum (no. of bronchodilators per day during run-in), geographical region, visit by baseline score and visit by treatment interactions included as covariates.
- Model using proc glimmax with; random visit / subject=subject\*period residual type=un statement to account for repeated visit;
- For TDI the model will use BDI in place of baseline score.
- For E-RS the model will use 4 weekly period in place of visit.
- This analysis will include all subjects with a non-missing baseline assessment.
   See Section 10.6.2.3 for details on how to handle missing data.

#### **Model Checking & Diagnostics**

UMEC will be used as the reference level for treatment for the comparison between UMEC/VI vs. UMEC. Salmeterol will be used as the reference level for treatment for the comparison between UMEC/VI vs. Salmeterol and UMEC vs Salmeterol.

## Secondary Statistical Analysis

 Pearson residuals will be plotted by using PLOTS=RESIDUALPANEL option for the model statement in SAS.

#### **Model Results Presentation**

• The odds ratio, 95% CI and p-value will be presented for UMEC/VI versus UMEC, UMEC/VI versus Salmeterol and UMEC versus Salmeterol.

## **Summary Results Presentation**

• The number and percentage of responders and non-responders at each visit will be summarized on the same table as the analysis results details above.

## Sensitivity and Supportive Statistical Analyses

• If the model fails to converge then the analyses will be carried out separately for each visit or 4 weekly period instead.

#### **COPD Exacerbation**

## **Secondary Statistical Analysis**

#### **Endpoints**

- Time to first on-treatment mild/moderate/severe COPD exacerbation
- Time to first on-treatment moderate/severe COPD exacerbation
- Time to first on-treatment severe COPD exacerbation

## **Model Specification**

• Cox's proportional hazards model,

#### Terms in the model:

Dependent variable: time to first on-treatment mild/moderate/severe exacerbation or moderate/severe exacerbation or severe exacerbation

Categorical: treatment group, stratum (no. of bronchodilators per day during run-in) and geographical region.

• Use the 'exact' method for handling ties. (If the analysis will not run using the 'exact' method, then the 'Efron' method for handling ties will be used instead.)

## **Model Checking & Diagnostics**

- The proportional hazards assumption for this method of analysis will be examined by obtaining the Kaplan-Meier estimates of the survival function S(t) over time separately for treatment group. Under the assumption of proportional hazard between the treatment groups, In{-In[S(t)]} for the two groups should be parallel to each other and the distance between them constant. If the curves are approximately parallel, then the proportional hazard assumption is not violated. If these curves cross each other or diverge greatly from the assumption of parallel lines, then the assumption is not met.
  - If model fails to converge, model will be investigated excluding the geographical region covariate.

## **Secondary Statistical Analysis**

#### **Model Results Presentation**

The Hazard ratio, 95% CI and p-value will be presented for comparison between UMEC/VI versus UMEC, UMEC/VI versus Salmeterol and UMEC versus Salmeterol.

## **Secondary Statistical Analysis**

## **Endpoints**

- Time to first on-treatment mild/moderate/severe COPD exacerbation
- Time to first on-treatment moderate/severe COPD exacerbation
- Time to first on-treatment severe COPD exacerbation

## **Model Specification**

 A Kaplan-Meier analysis will also be performed for figure showing Kaplan-Meier survivor functions of the proportion of subjects with a first exacerbation over time for each treatment group separately plotted on the same figure.

#### **Model Results Presentation**

- Probability of having an event, 95% CI and first quartile time to exacerbation (estimate of the time at which 25% of subjects in each treatment group would have had an exacerbation)
- Figure showing Kaplan-Meier survivor functions of the proportion of subjects with a first exacerbation over time for each treatment group separately plotted on the same figure.

#### CID

## **Secondary Statistical Analysis**

#### **Endpoints**

- Time to first deterioration of each of the individual components i.e. Trough FEV1, SGRQ total score, CAT score, TDI focal score
- Time to first CID composite endpoint (SGRQ, FEV1, EXAC (mod/sev))
- Time to first CID composite endpoint (CAT, FEV1, EXAC (mod/sev) )
- Time to first CID composite endpoint (CAT, SGRQ, TDI, EXAC (mod/sev) )

#### **Model Specification**

Cox's proportional hazards model,

## Terms in the model:

Dependent variable: time to endpoint of interest

Categorical: treatment group, stratum (no. of bronchodilators per day during run-in) and geographical region and respective baselines (i.e. endpoint includes CAT and SGRQ then include baselines for these 2 variables).

• Use the 'exact' method for handling ties. (If the analysis will not run using the 'exact' method, then the 'Efron' method for handling ties will be used instead.)

## **Model Checking & Diagnostics**

• The proportional hazards assumption for this method of analysis will be examined by obtaining the Kaplan-Meier estimates of the survival function S(t) over time separately for treatment group. Under the assumption of proportional hazard between the treatment groups, ln{-ln[S(t)]} for the two groups should be parallel to each other and the distance between them constant. If the curves are approximately parallel, then the proportional hazard assumption is

## **Secondary Statistical Analysis**

not violated. If these curves cross each other or diverge greatly from the assumption of parallel lines, then the assumption is not met.

#### **Model Results Presentation**

• The Hazard ratio, 95% CI and p-value will be presented for comparison between UMEC/VI versus UMEC, UMEC/VI versus Salmeterol and UMEC versus Salmeterol.

## **Summary Results Presentation**

 The total number of deteriorations (Yes/No) for each of the composite and the individual components for each treatment will be summarised. This will be produced for three the composite endpoint definitions.

## **Secondary Statistical Analysis**

#### **Endpoints**

- Time to first CID composite endpoint (SGRQ, FEV1, EXAC (mod/sev) )
- Time to first CID composite endpoint (CAT, FEV1, EXAC (mod/sev) )
- Time to first CID composite endpoint (CAT, SGRQ, TDI, EXAC (mod/sev))

#### **Model Specification**

 Kaplan-Meier survivor functions of the proportion of subjects with deterioration (composite and individual components) over time will be obtained for each treatment group separately and will be plotted on the same figure.

#### **Model Results Presentation**

- Probability of having an event, 95% CI and first quartile time to CID composite endpoint (estimate of the time at which 25% of subjects in each treatment group would have had a deterioration)
- Figure showing Kaplan-Meier survivor functions of the proportion of subjects with a first deterioration over time for each treatment group separately plotted on the same figure.

#### **Summary Results Presentation**

• The first quartile time to first deterioration (taken from the Kaplan Meier analysis) will also be presented in a summary table.

#### **Rescue Medication**

## **Secondary Statistical Analysis**

#### **Endpoints**

- Mean number of inhalations of rescue use per day (using eDiary)
- Percentage of rescue-free days (using eDiary)

## Model Specification, Checking and Results Presentation

- Similar to trough FEV1 in Section 7.1.5.1 where Visit is replaced with 4-weekly period.
- The model will use all available values:
  - Periods defined as Weeks 1-4, 5-8, 9-12, and up to Weeks 21-24
- Baseline is defined in Section 5.2
- Model will include the period by baseline and period by treatment interaction.
- Overall treatment effect from the same model using overall main effect on Lsmean statement.

## Sensitivity and Supportive Statistical Analyses

If the assumption of normality for the percentage of rescue-free days is not satisfied, a non-

## **Secondary Statistical Analysis**

parametric analysis of percentage of rescue-free days will be carried out. Hodges Lehman estimates for the median treatment difference and 95% CI based upon a Wilcoxon rank sum test will be used. The p-value will be based on Van Elteren test, an extension to the Wilcoxon rank sum test for two group comparison, stratified by geographical region.

## Trough FEV1, FVC and IC

## **Secondary Statistical Analysis**

#### **Endpoints**

- Ratio of trough FEV1 to baseline FEV1
- Trough FVC
- Trough IC

## **Model Specification**

- Ratio of trough FEV1 to baseline FEV1 at Week 24 will be analysed for the ITT population using a mixed model repeated measures (MMRM) including data recorded at each of Week 4, Week 12 and Week 24. The model will have a response of log (Trough FEV1/Baseline FEV1) with covariates of log (baseline FEV1), geographical region, stratum (no. of bronchodilators per day during run-in), visit, treatment, visit by log (baseline FEV1) and visit by treatment interactions, where visit is nominal. Results will be back transformed to provide point estimates for the ratios.
- Trough FVC and Trough IC endpoints above will be analyzed using the same methodology as the primary analysis of trough FEV1 (detailed in Section 7.1) using all available FVC or IC data recorded at Weeks 4, 12 and 24 and with relevant baseline. Baseline defined in Section 5.2.

The following will apply for all the endpoints FEV1, FVC and IC:

- The Kenward and Roger method (KR) for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- In the event the model fails to run using the KR method, then the residual method will be used instead.
- An unstructured covariance structure for the R matrix will be used by specifying 'type='UN'
  on the REPEATED line.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied but appropriate adjustments may be made based on the data.
- Normality assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the
  fitted values (i.e. checking the normality assumption and constant variance assumption of
  the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

Least squares (LS) mean and LS mean changes from baseline with their corresponding

## **Secondary Statistical Analysis**

standard errors (SEs) will be presented for each treatment by visit, together with estimated treatment differences (UMEC/VI 62.5/25 vs. UMEC 62.5, UMEC/VI 62.5/25 vs Salmeterol and UMEC 62.5 vs Salmeterol), corresponding 95% CIs and p-values.

- A plot of LS mean changes from baseline and 95% CIs for each treatment by visit will be generated.
- A plot of LS mean treatment differences and 95% CIs between the treatment groups by visit will also be generated.

## **Summary Results Presentation**

- Summary of baseline FVC will be presented by treatment for all subjects.
- Summary statistics for raw and change from baseline in trough FVC at each visit and for each treatment will be presented on the same table.
- Summary of baseline IC will be presented by treatment for all subjects.
- Summary statistics for raw and change from baseline in trough IC at each visit and for each treatment will be presented on the same table.

## **Subject Global Ratings of Change**

## **Secondary Statistical Analysis**

## **Endpoints**

- Subject global rating of COPD severity
- Subject global rating of change in COPD Severity

## **Model Specification**

 Change of Severity will be analyzed using a generalized linear mixed model with treatment as an explanatory variable and visit, stratum (no. of bronchodilators per day during run-in), geographical region, visit by treatment interactions included as covariates.

#### **Model Checking**

 Pearson residuals will be plotted by using PLOTS=RESIDUALPANEL option for the model statement in SAS..

#### **Model Results Presentation**

- Number and percentage of subjects reporting each category of change at each visit
- P-value for comparison between UMEC/VI 62.5/25 vs. UMEC 62.5, UMEC/VI 62.5/25 vs.
   Salmeterol and UMEC 62.5 vs. Salmeterol for change.
- UMEC will be used as the reference level for treatment for the comparison between UMEC/VI vs. UMEC. Salmeterol will be used as the reference level for treatment for the comparison between UMEC/VI vs. Salmeterol and UMEC vs Salmeterol.

## 7.3. Exploratory Efficacy Analyses

## 7.3.1. Endpoint / Variables

- 1) Annual rate of on-treatment mild/moderate/severe exacerbations
- 2) Annual rate of on-treatment moderate/severe exacerbations
- 3) Mean number of inhalations of rescue use per day (using eMDI)
- 4) Percentage of rescue-free days (using eMDI)
- 5) To compare physical activity levels, ER-S, rescue medication use, exacerbations and mortality in subjects with and without a CID
- 6) Physical activity

## 7.3.2. Summary Measure

- 1) Rate ratio
- 2) Rate ratio
- 3) Mean change from baseline
- 4) Mean change from baseline
- 5) Mean change from baseline
- 6) Mean change from baseline

## 7.3.3. Population of Interest

The exploratory analyses will be based on the ITT population apart from the physical activity endpoint and deterioration status at 24 weeks to predict the outcome of physical activity levels, which will be based on the AM population.

## 7.3.4. Strategy for Intercurrent (Post-Randomization) Events

• All Endpoints will use the same strategy for intercurrent events as defined in Section 7.1.4.

# 7.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.3.5.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

#### 7.3.5.1. Statistical Methodology Specification

#### **Exploratory Statistical Analyses**

#### **Endpoints**

- Annual rate of on-treatment mild/moderate/severe exacerbations
- Annual rate of on-treatment moderate/severe exacerbations

#### **Model Specification**

Generalized linear model assuming a negative binomial distribution,

## **Exploratory Statistical Analyses**

#### Terms in the model:

Response: number of on-treatment mild/moderate/severe exacerbations or moderate/severe exacerbations per subject

Categorical: treatment group, exacerbation history ( $\leq 1, \geq 2$  of severity endpoint), stratum (no. of bronchodilators per day during run-in) and geographical region.

Offset: logarithm of time on treatment

## **Model Checking & Diagnostics**

- The fit of the regression models will be examined using "Q-Q" plots of the standardized residuals. Interpretation of these plots will be aided by the addition of simulated envelopes as proposed by Atkinson (Atkinson, 1985). Should the model not fit with all specified covariates (fixed effects with very large estimates/variances) then geographical region will be dropped from the model.
- If there are concerns over model fit then an over dispersed poisson model will be investigated.

#### **Model Results Presentation**

Treatment group mean annual exacerbation rates, treatment rate ratio and associated 95% CI will be presented and p-values will be presented.

Analysis is limited by number of moderate and severe exacerbations possible before withdrawal to the study and due the assumption they continue at this rate post withdrawal. Output to be appropriately footnoted.

# **Exploratory Efficacy Statistical Analyses**

## **Endpoints**

- Mean number of occurrences of rescue use per day (using eMDI)
- Percentage of rescue-free days (using eMDI)

## Model Specification, Checking and Results Presentation

- Similar to trough FEV1 in Section 7.1.5.1 excluding visit from the model
  - Baseline is defined in Section 5.2

#### **Exploratory Statistical Analyses**

## **Endpoints**

- Deterioration Status at Day 30 to predict short term outcomes:
  - o ER-S
  - Rescue medication use (Mean number of inhalations of rescue use per day (using eDiary))
  - Mortality
  - Hospitalised Exacerbations

#### Model Specification

 Change in E-RS and mean number of inhalations of rescue use per day will be compared between subjects who have and have not experienced deterioration up to and including day 30, using a MMRM model. The following covariates will be included in the model: treatment,

## **Exploratory Statistical Analyses**

deterioration status at day 30, baseline, geographical region, stratum (no. of bronchodilators per day during run-in), 4-weekly period, deterioration status at day 30 weeks by 4 weekly period, and 4-weekly period by baseline interactions. Data will only be included post visit 3.

• The time to first hospitalized exacerbation after day 30 and time to mortality after day 30 will be presented for subjects with and without deterioration at day 30. The actual time to post day 30 hospitalised exacerbation and mortality will be analysed using a Cox's proportional hazards models, with covariates treatment group, stratum (no. of bronchodilators per day during run-in) and geographical region, and deterioration at day 30.

## **Model Checking & Diagnostics**

- The Kenward and Roger method (KR) for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used. In the event the model fails to run using the KR method, then the residual method will be used instead.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the
  fitted values (i.e. checking the normality assumption and constant variance assumption of
  the model respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

- For E-RS and mean number of inhalations of rescue use per day the adjusted means, pairwise differences, p-values and 95% confidence limits for the deterioration status differences will be summarised at visit 4 and visit 5 only.
- For mortality and hospitalized exacerbations, the Hazard ratio, 95% CI and p-value will be presented for the comparison between deterioration status.

## **Summary Results Presentation**

 A summary of subjects who have and have not experienced a first deterioration at day 30 will be presented.

#### **Exploratory Statistical Analyses**

#### **Endpoints**

Physical activity

- Change from baseline in step count
- Change from baseline in light activity duration
- Change from baseline in moderate to vigorous physical activity duration
- Change from baseline in total energy expenditure

#### **Model Specification**

- The dataset containing the mean value for each subject-visit will be used to look at differences between baseline, Week 1, Week 4 and Week 24.
- MMRM will be used to model each activity variable against the treatment group variable including data recorded at each of baseline, Week 1, Week 4 and Week 24.

• Other covariates included will be the mean of the activity monitor variable at baseline and smoking status.

## **Model Checking**

• The physical activity endpoints will be plotted in histograms to view their distributions and enable possible sensitivity analyses.

#### **Model Results Presentation**

• Estimated mean change from baseline for each treatment group will be calculated from the model and displayed with their associated standard errors. The estimated treatment difference will also be presented together with 95% confidence intervals (CIs) for the difference and p-value.

## **Summary Results Presentation**

• Summaries will include the means and standard deviations of the activity monitor variables at the four time points by treatment group.

## **Sensitivity and Supportive Statistical Analyses**

• If the histogram for change in step count or light activity duration or moderate to vigorous physical activity duration or total energy expenditure is not normally distributed, a transformation of the variable may be considered. If the MMRM analysis shows that the model is ill-fitting then a Mann-Whitney test (non-parametric t-test) will be used to look at the change in activity monitor outputs between each treatment group at Week 1, Week 4 and Week 24.

# 7.4. Subgroup Analyses

# **Subgroup Analysis**

## **Endpoints**

Repeat specified analyses/displays for:

- Study Population
- Efficacy
- Safety

Output for subgroup analysis indicated in Section 10.8.8

# Model Specification

• Analysis will be performed 'by' each subgroup separately. Please refer to main endpoint model for model specification.

# **Model Checking & Diagnostics**

• As per main endpoint

# **Model Results Presentation**

• As per main endpoint

## 8. SAFETY ANALYSES

The safety analyses will be based on the ITT population, unless otherwise specified. Data collected after completion or withdrawal of study treatment will be considered post-treatment and included in relevant displays.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

The 10 most frequent on-treatment adverse events in each treatment will be summarised. In case of ties in frequency all AEs for that frequency will be displayed. On-treatment AEs experienced by 3 % (without rounding) or more of subjects in any treatment group will also be displayed. The most common on-treatment serious drug-related and most common on-treatment non-serious drug-related adverse events will be based on events experienced by 3% (without rounding) or more of subjects in any treatment group.

Classification of an AE as pre-, on- or post-treatment is provided in Section 10.3.2. All listings of AEs/SAEs will include an identification of the treatment phase (see Section 10.3.2).

## 8.2. Adverse Events of Special Interest Analyses

Adverse events (AEs) of special interest (AESI) have been defined as AEs which have specified areas of interest for UMEC, VI or for the COPD population. A list of Standardized Medical Dictionary for Regulatory Affairs (MedDRA) Queries (SMQs) and other groupings for AESI is provided in Section 10.5.4.

Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the planned displays are provided in Appendix 8: List of Data Displays.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations for liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 8: List of Data Displays.

## 9. REFERENCES

Atkinson, AC. (1985) Plots, Transformations and Regression. Clarendon Press.

Evidera. (2013). E-RS (EXACT-Respiratory Symptoms (Version 2.0). Bethesda, MD: Author.

GlaxoSmithKline Document Number 2016N277425\_00 Study ID 201749. (A 24-week treatment, multi-center, randomized, double-blind, double-dummy, parallel group study to compare Umeclidinium/Vilanterol, Umeclidinium, and Salmeterol in subjects with chronic obstructive pulmonary disease (COPD) Report Date 13-SEP- 2016.

GOLD. Global Initiative for Chronic Obstructive Lung Disease (Updated 2018). http://www.goldcopd.org.

Jones, St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Manual. March 2016 (Version No. 1.3)

Ratitch, B., O'Kelly, M. and Tosiello, R. (2013), Missing data in clinical trials: from clinical assumptions to statistical analysis using pattern mixture models. Pharmaceut. Statist., 12: 337–347. doi: 10.1002/pst.1549
# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

# 10.1.1. Protocol Defined Schedule of Events

| Visit<br>Week | Pre-<br>screen <sup>1</sup><br>0<br>-10 to -4 | Screen/<br>Run-in<br>1 | Rando-<br>mization<br>2 | Blinded<br>3<br>4 | Treatment 4 12 | 5<br>24 | EW<br>Visit <sup>2</sup> | Telephone Follow up contact 6 |
|---|---|---|---|---|---|---|---|---|
| Day | -70 to -28 | -28 | 1 | 28 | 84 | 168 | | 7 days after V5 or EW<br>Visit |
| Window | -7/+2 days | -7/+2 days | -7/+2<br>days | -7/+2 days | -7/+2 days | -7/+2 days | | ±3 days |
| Screen/Baseline | | | | | | | | |
| Informed consent | Х | | | | | | | |
| Demography | Х | | | | | | | |
| Medical/COPD history | | Х | | | | | | |
| Smoking history/status | | Х | | | | | | |
| Smoking cessation counselling | | Х | | | | | | |
| Concomitant medication assessment | Х | Χ | Χ | Х | Х | Х | X | X |
| Height and weight | | Χ | | | | | | |
| Cardiovascular History/family history of premature CV disease]) | | X | | | | | | |
| Screening spirometry (including post bronchodilator testing) <sup>3</sup> | | Х | | | | | | |
| CAT questionnaire | | Х | Χ | | | | | |
| Verify Inclusion/Exclusion Criteria | | Х | | | | | | |
| Training on use of inhalers | | Х | Х | | | | | |
| Training on use of eDiary and eMDI | | Х | Х | | | | | |
| Verify randomization Criteria | _ | | Х | _ | _ | | | |

| | | | | Rlinded | Treatment | | EW<br>Visit <sup>2</sup> | Telephone Follow up contact 6 7 days after V5 or EW Visit ±3 days |
|---|---|---|---|---|---|---|---|---|
| Visit<br>Week | Pre-<br>screen <sup>1</sup><br>0<br>-10 to -4 | Screen/<br>Run-in<br>1 | Rando-<br>mization<br>2<br>0<br>1<br>-7/+2<br>days | 3 4 | 4 12 | 5<br>24 | | |
| Day | -70 to -28 | -28 | | 28 | 84<br>-7/+2 days | 168<br>-7/+2 days | | |
| Window | -7/+2 days | -7/+2 days | | -7/+2 days | | | | |
| Register Visit in InForm | X | Х | Х | Х | Х | Х | Х | X |
| Register Visit in RAMOS NG | Х | Х | Х | Х | Х | Х | Х | X |
| Efficacy/HRQoL assessments | | | | | | | | |
| Spirometry, including pre-dose FEV <sub>1</sub> , trough FEV <sub>1</sub> and inspiratory capacity | | | Х | Х | Х | Х | | |
| SAC BDI questionnaire 4 | | | Х | | | | | |
| SAC TDI questionnaire <sup>4</sup> | | | | Х | Х | Х | | |
| SGRQ-C questionnaire <sup>4</sup> | | | Х | Х | Х | Х | | |
| CAT questionnaire 4 | | Χ | Х | Χ | Χ | Χ | | |
| EXACT/ER-S: COPD 5 | | | | | | <b>→</b> | | |
| Patient Global Rating of COPD severity | | | Х | Х | Х | Χ | | |
| Patient Global Rating of Change in COPD | | | | Х | Х | Х | | |
| Safety assessments | | | | | | | | |
| Adverse events/Serious adverse events 6 | Х | X | Χ | X | X | Χ | Х | Χ |
| COPD exacerbation assessment | Х | Х | Х | Х | Х | X | Х | Х |
| 12-Lead ECG | | X | | | | | | |
| Urine pregnancy test <sup>7</sup> | | X | Х | | | Χ | Х | |
| Pharmacogenetic sample <sup>8</sup> | | | lacksquare | | Х | | <u> </u> | |
| Medication/Supplies | | | T | 1 | r | | | 1 |
| Dispense rescue albuterol/slabutamol. Dispense MDI <sup>9</sup> | | Х | X | Х | Х | Х | | |
| Assess COPD medication compliance <sup>10</sup> during run-in | | ,, | Х | | | | | |
| Dispense eDiary | | Х | | | | | | |
| Assess compliance with eDiary during run-in | | | X | | | | V | |
| Collect rescue albuterol/slabutamol. | | | X | X | X | Χ | Χ | |

| Visit Week Day Window | Pre-<br>screen¹<br>0<br>-10 to -4<br>-70 to -28<br>-7/+2 days | Screen/<br>Run-in<br>1<br>-4<br>-28 | Rando-<br>mization<br>2<br>0<br>1<br>-7/+2<br>days | 3<br>4<br>28<br>-7/+2 days | 12<br>84<br>-7/+2 days | 5<br>24<br>168<br>-7/+2 days | EW<br>Visit <sup>2</sup> | Telephone Follow up contact 6 7 days after V5 or EW Visit ±3 days |
|---|---|---|---|---|---|---|---|---|
| Collect eDiary | | | | | | Х | Х | |
| Dispense study treatment <sup>11</sup> | | | Χ | Х | Х | | | |
| Collect study treatment | | | | X | X | Χ | Χ | |
| Assess study treatment compliance during treatment <sup>10</sup> | | | | X | Х | Χ | Х | |
| Study sub-set | | | | | | | | |
| Physical activity monitor <sup>12</sup> | | Х | Χ | X | | Χ | | |
| Collect Physical activity monitor | | | | | | Χ | Χ | |

- 1. Pre-screen Visit 0 must be completed prior to Screening Visit1. It can be completed 6 weeks prior or on the same day of V1, if no wash out of exclusionary medications is required.
- 2. Early Withdrawal Visit: Subjects that withdraw should return to the clinic as soon as possible to complete the Early Withdrawal Visit procedures.
- 3. Spirometry at screening should be performed as described in (Section 7.2.2.1 in the protocol).
- 4. SAC BDI, SAC TDI, SGRQ-C, CAT questionnaires will be completed at clinic visits and in the eDiary
- 5. EXACT/ER-S: COPD is completed daily in the eDiary approximately 2 hours before bed-time, starting on Day 1 of the run-in period.
- 6. For the start date of collecting AEs and SAEs see (Appendix 4)
- 7. Pregnancy test: for females for child bearing potential only.
- 8. Pharmacogenetic sample may be drawn at visit 2 or any visit after.
- 9. Rescue medication use to be recorded in the eDiary daily and in some sites in the eDiary and the eMDI
- 10. Sites are requested to call subjects every 2 weeks to remind them to take study treatment regularly and to record the time of the morning and evening dose in the eDiary.
- 11. In order to ensure subjects have sufficient doses of study treatment, they must return to clinic within 30 days from V2 and within 60 days from V3 respectively.
- 12. The Actigraph GT9X should be worn for 7 days from Visit 1, for 7 days from Visit 2, for 7 days from Visit 3 and for 7 days prior to Visit 5.

# 10.2. Appendix 2: Assessment Windows

# 10.2.1. Definitions of Assessment Windows for Analyses

Data are generally reported according to the nominal time of clinic visits and assessments as specified in the protocol, and time windows for exclusion will not be defined. For example, if a subject recorded values for the Week 4 (Day 28) visit that were actually made on the 21st day of treatment, they will be presented as Week 4 (Day 28) values in the summary tables.

# 10.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 10.3.1. Study Phases for Concomitant Medication

The following rules will be used to classify a concomitant medication as being taken during one or more study treatment phases (pre-treatment, on-treatment and post-treatment):

| | Definition | | |
|---|---|---|---|
| Study Phase | Pre-<br>Treatment | On-<br>Treatment | Post-<br>Treatmen<br>t |
| Subject did not take study treatment (e.g, screen failures) and conmed stop date > date of Screening or variable that asks if conmed is on-going (refer hereafter as goingmed) is "yes" | Y | | |
| (Conmed start date <treatment (refer="" <="" and="" as="" asks="" conmed="" date="" date<="" hereafter="" if="" is"="" medication="" of="" or="" prior="" priormed))="" screening="" start="" stop="" study="" taken="" td="" that="" to="" treatment="" variable="" yes"=""><td>Y</td><td></td><td></td></treatment> | Y | | |
| (Conmed start date <treatment and="" conmed="" date="" date<="" is="" or="" priormed="" start="" stop="" td="" treatment="" yes)="" ≤=""><td>Y</td><td>Y</td><td></td></treatment> | Y | Y | |
| (Conmed start date <treatment (conmed="" and="" date="" is="" or="" priormed="" start="" stop="" yes)="">treatment stop date or goingmed is "yes")</treatment> | Y | Y | Y |
| (Treatment start date ≤ conmed start date <treatment stop<br="">date and treatment start date ≤ conmed stop date ≤<br/>treatment stop date) or (Treatment start date=conmed start<br/>date=conmed stop date=treatment stop date)</treatment> | | Y | |
| ([Treatment start date ≤ conmed start date <treatment (conmed="" [treatment="" and="" date="" date]="" date])="" or="" start="" stop="">treatment stop date or goingmed is Yes)</treatment> | | Y | Y |
| Conmed start ≥ treatment stop date and treatment start date<br>≠ treatment stop date | | | Υ |

#### 1. NOTES:

- The duration of a single concomitant medication can extend over multiple study phases
- Please refer to Appendix 6: Reporting Standards for Missing Data for handling of partial dates for concomitant medication.
- Note: If priormed or goingmed flags are missing or inconsistent, then medications will be assigned to all applicable phases.

# 10.3.2. Study Phases for Adverse Events and All Other Data Recorded in Logs (excluding Concomitant Medications)

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date + 1 |

# 10.3.3. Treatment Emergent Flag for Adverse Events and Exacerbations

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop date plus one day.</li> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 1.</li> </ul> |

# NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

# 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | Reporting Area |
| HARP Server | : uk1salx00175 |
| HARP Compound : gsk573719_gw642444/mid201749/final | |
| Analysis Datasets | |

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.0 or higher].
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all tables in the final reporting effort for use in writing the CSR.

### 10.4.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the randomised treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - FEV<sub>1</sub>, FVC and IC will have a min and max to 2dp and then follow IDSL standards to reporting other summary statistics
  - SGRQ and TDI will have a min and max to 1dp and then follow IDSL standards to reporting other summary statistics
  - CAT will have a min and max to 0dp and then follow IDSL standards to reporting other summary statistics
  - Odds Ratios and Hazard Ratios will be reported to 2dp

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated. Actual time will be used for calculation of times to events and Kaplan-Meier plots.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will only be included in summary tables as part of 'minimum/maximum post baseline' and 'minimum/maximum change from baseline' summary.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | Categorical Data N, n, frequency, % |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

### **Study Day**

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < treatment start date → Study Day = Ref Date treatment start date
- Ref Date ≥ treatment start date → Study Day = Ref Date (treatment start date) + 1

# Completer

A study completer will be defined as a subject who completes the visit 5 trough FEV1
assessment.

# 10.5.2. Study Population

# **Demographics**

# Age

- Since the eCRF only collects the year of birth, GSK standard IDSL algorithms will be used for calculating age where date and month will be imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated based on the Pre-screening visit date.

# Age Category

- Age categories are based on age at Pre-screening and are defined as:
  - ≤64 years
  - 65-74 years
  - 75-84 years
  - ≥85 years

# **Body Mass Index (BMI)**

• Calculated as Weight (kg) / Height (m)<sup>2</sup>

## **Smoking Status**

Smoking status at Screening is determined directly from the eCRF.

#### **Maintenance Naive/Non Maintenance Naive**

 Maintenance naive (MN) is defined as subjects with no COPD maintenance medication apart from short-acting bronchodilators recorded in the 30 days prior to screening (evaluation period 30 days prior to screening until 1st study treatment).

### **Reversibility and GOLD Classifications**

### Reversibility

- A subject's responsiveness to salbutamol at Screening will be classified as 'Reversible' or 'Nonreversible' based on the difference between their pre-salbutamol assessment of FEV<sub>1</sub> and their post-salbutamol assessment of FEV<sub>1</sub> as follows:
  - Reversible, if they had a difference in FEV1 of ≥ 12 % and ≥ 200 mL, or
  - Non-reversible, if they had a difference in FEV1 of < 200 mL or a ≥ 200 mL difference that was < 12 % of the pre-salbutamol FEV1.

#### **GOLD Grade 1-4**

Based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2018), Subjects will be classified into GOLD Grades 1-4 using the post-salbutamol percent predicted FEV<sub>1</sub> assessment at Screening (Visit 1):

- GOLD Grade 1 (Mild): Percent Predicted FEV<sub>1</sub> ≥ 80%
- GOLD Grade 2 (Moderate): 50% ≤ Percent Predicted FEV<sub>1</sub> < 80%</li>
- GOLD Grade 3 (Severe): 30% ≤ Percent Predicted FEV<sub>1</sub> < 50%</li>
- GOLD Grade 4 (Very Severe): Percent Predicted FEV<sub>1</sub> < 30%</li>

# **GOLD Category A-D (Using CAT)**

GOLD (CAT) Category A-D definitions as follows:

- A. Low risk, less symptoms: CAT < 10; ≤1 moderate exacerbation; and no hospitalizations for exacerbations, prior year.
- B. Low risk, more symptoms: CAT ≥ 10; ≤1 moderate exacerbation and no hospitalizations for exacerbations, prior year
- C. High risk, less symptoms: CAT < 10; ≥ 2 moderate exacerbations, prior year OR >=1 leading to COPD hospitalization, prior year
- D. High risk, more symptoms: CAT ≥ 10; ≥ 2 moderate exacerbations, prior year OR >=1 leading COPD hospitalization, prior year

#### Long-acting Bronchodilator Usage During the Run-in (Randomisation Stratum)

Randomization stratum, long-acting bronchodilator usage during the run-in, will be derived based on the RMC classification and will be grouped into the following 2 categories:

- None
- One long-acting bronchodilator per day

Long-acting bronchodilator is defined as any COPD medication in Respiratory Medication Class (MRC) under 'Long-acting beta-2 agonist – Group 2' or 'Long-acting beta-2 agonist – Group 3' or 'Long-acting anticholinergic'.

Randomisation stratum is also collected at randomization in RAMOS NG and on eCRF. All randomisation stratum (RANDALL NG, eCRF and derived) will be listed.

### Compliance

# **ELLIPTA DPI Compliance**

The number of doses of study treatment taken by each subject from each inhaler will be calculated from the dose counter start and stop counts for each inhaler used. If a dose counter start count is missing then it will be assumed to be 30. If all dose counter stop counts are non-missing then the percentage compliance will be calculated as:

Compliance = <u>sum of all (dose counter start – dose counter stop) x 100</u> (exposure stop date – exposure start date +1)

- If any dose counter stop is missing then the treatment compliance will be set to missing for that subject.
- If the dose counter start=dose counter stop then it will be assumed that no doses were taken from that container.

# **DISKUS Compliance**

The number of doses of study treatment taken by each subject from each inhaler will be calculated from the dose counter start and stop counts for each inhaler used. If a dose counter start count is missing then it will be assumed to be 60. If all dose counter stop counts are non-missing then the percentage compliance will be calculated as:

Compliance = <u>sum of all (capsules dispensed –capsules returned) x 100</u> 2 x (exposure stop date – exposure start date +1)

 If any dose counter stop is missing then the treatment compliance will be set to missing for that subject.

# **Overall Compliance**

- The average of the compliance with the ELLIPTA DPI and compliance with the DISKUS. If the
  compliance with any of the two inhalers is missing then the overall compliance for that subject
  will be considered missing.
- Overall compliance and compliance with each type of inhaler will be categorised as follows:
  - < 80 %
  - $\geq$  80 % to < 95 %
  - ≥ 95 % to ≤105 %
  - >105 % to ≤120 %
  - >120 %.
- If a subject received a treatment other than the randomized treatment during the study, the compliance will still be calculated using data from all containers received and overall exposure start and stop dates.

#### **Cardiovascular Risk Factors**

 Subjects with at least one of the following current or past medical conditions at Screening will be classed as having a cardiovascular (CV) risk factor. The number of CV risk factors at Screening (0, 1, or >=2) will be derived.

#### Cardiovascular Risk Factors

- Coronary artery disease
- Myocardial infarction
- Arrhythmia
- Congestive heart failure
- Hypertension
- Cerebrovascular accident
- Diabetes mellitus
- Hypercholesterolemia

### **Concomitant Medications and COPD Exacerbation History**

#### **COPD Concomitant medications**

COPD concomitant medications given for an exacerbation will be grouped into the following RMCs based on pre-defined code lists derived from ATC classifications:

- Androgens and Estrogens
- Anti-IgE, Anti-IL5
- Anticholinergic
- Antiinfectives (antibiotics, antiseptics)
- Antimycotics
- Antivirals
- Short-acting anticholinergic
- Short-acting beta-2 agonist
- Long-acting anticholinergic
- Long-acting beta-2 agonist
- Xanthine
- PDE4 Inhibitors
- Corticosteroid inhaled
- Corticosteroid depot
- Corticosteroid systemic oral parenteral and intra-articular
- Corticosteroid other
- Leukotriene receptor antagonist
- Nedocromil or cromolyn sodium
- Mucolytics
- Oxygen
- Other medication given for exacerbation
- Other COPD medication

# **COPD Exacerbation History**

- Number of COPD exacerbations reported in the past year prior to Screening will be summarised (0, 1, =>2) according to the following categories: mild COPD exacerbation, moderate COPD exacerbation, severe COPD exacerbation, mild/moderate/severe COPD exacerbation, moderate/severe COPD exacerbation and severe COPD exacerbation.
- Moderate COPD exacerbations are defined as exacerbation that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalisation).
- Severe COPD exacerbations are defined as exacerbations that required in-patient hospitalisation.

### **Concomitant Medications and COPD Exacerbation History**

- Total number of mild/moderate/severe COPD exacerbations are defined as total numbers of mild, moderate and severe COPD exacerbation for each subject.
- Total number of moderate/severe COPD exacerbations are defined as total numbers of moderate and severe COPD exacerbation for each subject.

# **10.5.3.** Efficacy

#### **Spirometry**

Predicted FEV<sub>1</sub>, Absolute and Percent Reversibility in FEV<sub>1</sub>, Percent Predicted FEV<sub>1</sub> and Presalbutamol and Post-salbutamol FEV<sub>1</sub>/FVC Ratio

• These derived items will be delivered in a dataset from the vendor for central spirometry, except for post-salbutamol FEV<sub>1</sub>/FVC ratio, and no recalculation will be performed. Post-salbutamol FEV<sub>1</sub>/FVC ratio will be calculated as the ratio of post-salbutamol FEV<sub>1</sub> and FVC values.

### Trough

- The trough value for FEV<sub>1</sub>, FVC and IC at each of Weeks 4, 12 and 24 is calculated from the values at the assessments made 23 h and 24 h after dosing on the previous day.
- If the actual time of an assessment is after the time of dosing on the current day, the value for FEV<sub>1</sub>, FVC and IC will not be used in the calculation of trough.
- If one of the values is missing or excluded then the trough will be the single remaining value; otherwise the trough will be the mean of the two values.





#### CAT

#### **CAT Score**

- The CAT consists of eight items each formatted as a six-point differential scale: 0 (no impact) to 5 (high impact). A CAT score will be calculated by summing the non-missing scores on the eight items. The score can have values ranging from 0 to 40.
- If one item is missing, then the score for that item is set as the average of the non-missing items. If more than one item is missing, then the CAT score will be set to missing.
- If the language of the CAT conducted at a post-baseline visit is different to the language used at baseline, the CAT score for that visit and all subsequent visits will be set to missing.

# **CAT Responder**

- A subject will be considered a 'responder' according to CAT at each visit if their CAT score has
  decreased at least 2 units from baseline CAT score.
- A subject will be considered a 'non-responder' if their CAT score has decreased by less than 2
  units, has not changed or has increased compared to baseline.
- Missing data will be handled as detailed in Section 10.6.2.

#### **COPD Exacerbations**

#### General

- The duration of the exacerbation will be calculated as (exacerbation resolution date or date of death exacerbation onset date + 1).
- The time to the first on-treatment exacerbation will be calculated as (exacerbation onset date of first on-treatment exacerbation date of start of treatment + 1).
- For summaries/analyses, subjects will be represented from their Day 1 date to the start date of their first event up to and including their treatment stop date+1 day.
- Subjects that have not withdrawn from study treatment or experienced the event are censored

#### **COPD Exacerbations**

at their treatment stop date+1 day.

• The event rate for exacerbations will be lovemocalculated as the total number of events divided by the total annual subject exposure during the time-period of interest

### Severity

- Each COPD exacerbation will be categorized based on severity as follows:
  - Mild: no treatment with oral/systemic corticosteroids and/or antibiotics and no hospitalisation
  - Moderate: required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalisation).
  - Severe: required in-patient hospitalization or emergency room
  - Certain displays will include only moderate/severe exacerbations.

### **Calculation of Daily eDiary Endpoints**

#### General

Subjects were instructed to complete the daily eDiary in the evening (typically at bedtime). The parameters collected include rescue use and EXACT-PRO scores.

The table below shows which daily eDiary records are used to calculate the daily eDiary parameters for each period. Any diary data collected in the post-treatment phase of the study will not be slotted.

| Daily | Record | Analysis Time Period |
|---------------------------|---------------------------|----------------------|
| Beginning Timepoint (day) | Ending Timepoint<br>(day) | |
| -28 | -1 | Week -1 (Baseline) |
| 1 | 28 | Weeks 1 – 4 |
| 29 | 56 | Weeks 5 – 8 |
| 57 | 84 | Weeks 9 – 12 |
| 85 | 112 | Weeks 13 – 16 |
| 113 | 140 | Weeks 17 – 20 |
| 141 | 168 | Weeks 21 – 24 |
| 1 | 168 | Weeks 1 – 24 |

Note: There is no Day 0. Any records with actual day>168 will not be assigned to a time period. Note: Daily eDiary records that were not assigned to a time period will not be used in calculation of daily eDiary endpoints.

- For use of rescue medication endpoint, for a subject to be counted in a time period (except for baseline where at least 14 days non-missing entries required) they must have at least one diary entry recorded for that endpoint during that time period.
- For E-RS endpoint, for a subject to be counted in a time period they must have at least 16 days non-missing diary entries recorded for that endpoint during that time period.
- Any daily diary data that were collected post-study treatment discontinuation will be excluded from any analyses, including 4-weekly interval data summaries.

### Calculation of Daily eDiary Endpoints

# **Use of Rescue Medication via E-diary**

• The mean number of inhalations of rescue use per day and percentage of rescue-free days will be calculated during the 4-weekly interval intervals defined above.

#### **EXACT PRO**

### **EXACT Respiratory Symptoms**

 The 4-weekly mean scores for E-RS, and the subscales RS-Breathlessness, RS-Cough and Sputum, and RS-Chest Symptoms will be calculated as the mean of the daily scores in the 4weekly intervals defined above.

### **EXACT-RS** and Subscale Scores Responder

For each four weekly period;

- A subject will be considered as a responder according to E-RS total score if their 4- weekly mean change from baseline EXACT–RS ≤ -2.0.
- A subject will be considered as a non-responder according to E-RS total score if their 4-weekly mean change from baseline EXACT–RS >-2.0.
- A subject will be considered as a responder according to RS-Breathlessness score if their 4weekly mean change from baseline RS-Breathlessness ≤ -1.0.
- A subject will be considered as a non-responder according to RS-Breathlessness score if their 4-weekly mean change from baseline RS-Breathlessness >-1.0.
- A subject will be considered as a responder according to RS-Cough & Sputum score if their 4weekly mean change from baseline RS-Cough & Sputum ≤ -0.70.
- A subject will be considered as a non-responder according to RS-Cough & Sputum score if their 4-weekly mean change from baseline RS-Cough & Sputum >-0.70.
- A subject will be considered as a responder according to RS-Chest Symptoms score if their 4weekly mean change from baseline RS-Chest Symptoms ≤ -0.70.
- A subject will be considered as a non-responder according to RS-Chest Symptoms score if their 4-weekly mean change from baseline RS-Chest Symptoms >-0.70.
- Missing data will be handled as outlined in Section 10.6.2.

#### Rescue use for EMDI

- Will be analysed over Weeks 1 24 only
- The Medication Sensor Observation Period for each subject will be defined by the first date of sensor sync and the last date of sensor sync recorded in the database. Since a recorded rescue inhaler usage event in the database is also considered a sync event, if no first sync date is recorded, the date of the first rescue inhaler usage event will be used as the start date of observation. If no last sync date is recorded, the date of the last rescue inhaler usage event will be used as the end date of observation.
- A rescue occasion is defined as an inhaler usage event(s) in which one or more puffs occur within 2 minutes of each other, starting with the first reported puff.
- Days within the Medication Sensor Observation Period with no recorded rescue inhaler usage by the sensor will be assigned a rescue inhaler usage of 0.

#### Deterioration

- A Clinically Important Deterioration (CID) will be defined by a composite endpoint. A subject is
  considered to have deteriorated if, in the period from start of treatment to treatment stop + 1
  day, one or more of the following occurs (definition dependent);
- A decrease from baseline of ≥100mL in Trough pre-bronchodilator FEV1
- An increase from baseline of ≥4 units in SGRQ total score
- An exacerbation
- An increase from baseline of ≥2 units in CAT Score
- A TDI score of ≤-1 unit
- Subjects who are withdrawn from the study or have missing data will be included in analyses wherever possible. No imputation for missing data will be made.
- A subject [who had not met the deterioration definition at another timepoint] will be classed as not deteriorated and will be censored at their treatment stop date+1 day.
- To be evaluable for deterioration assessment you must have at least 1 post baseline assessment (not including exacerbations) for at least one of the individual components or had an exacerbation.
- For day 30 status assessment a subject will be classed as deteriorated if they had not met the
  deterioration definition by Day 30. To be evaluable for Day 30 deterioration status assessment
  you must have at least 1 post baseline assessment (not including exacerbations) for at least
  one of the individual components or had an exacerbation prior or on Day 30.

### **Physical Activity Monitoring**

- The data for Actigraph is generated as minute by minute for the amount of time worn on the body. The device generates the summary of each subject's daily total with the times the device was not worn excluded (WEAR - DAY TIME) and time not worn included (TOTAL - DAY TIME). The time that the device is worn is algorithmically detected. For analysis, we will only consider the daily summary data where the device was worn (WEAR - DAY TIME).
- For the physical activity monitoring analysis, a day will only be considered valid if the activity monitor is worn for at least 23 hours<sup>1</sup>. A minimum of 3 days<sup>2</sup> for each visit, visit 1 (baseline), visit 2 (randomization, week 1), visit 3 (week 4) and visit 5 (week 24), are needed in the analysis in order to have an accurate view of subjects' activity for each week. Only valid days within the 7 days after visit 1, after visit 2, after visit 3 and 7 days before visit 5 will be used in the primary analysis. Additional days may be used for further exploration of the data if deemed useful.
- To get a single observation per subject per visit, the mean of the daily values will be calculated for the week (no less than 3 days and no more than 7 days).
- Table 2.1 shows examples of acceptable and unacceptable weeks after visit 1 to use in the analysis. The boxes with an 'x' indicate days with valid activity monitor data. The day of the study visit will not be used since the activity may be out of the ordinary or not meet the minimum requirement of 23 hours. For instance, if a subject had visit 1 on January 1st, 2016, the acceptable days for use would be January 2nd to January 8th (Day 2 through 8) for a total of 7 days. Data from January 9th would not be used as it is out of scope of the week-long observation criteria. Examples of selection of days for visit 2, visit 3 and visit 5 are shown in Table 2.2, Table 2.3 and Table 2.4 respectively.

Table 2.1 Examples of Visit 1 Day Selection for Activity Monitor Analysis

| Days With Valid Activity Monitoring Data | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Day of Activity | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | Use/Do Not Use |
| Monitoring<br>Target Study<br>Day | Visit 1 | Study Day<br>-27 | Study Day<br>-26 | Study Day -<br>25 | Study Day<br>-24 | Study<br>Day -<br>23 | Study<br>Day -<br>22 | Study<br>Day -<br>21 | Study<br>Day -<br>20 | |
| Subject PP<br>Subject | X<br>X | X | X | X<br>X | X<br>X | X<br>X | x<br>x | X | X | Use Days 2-8<br>Use Days 4-8 |
| Subject | | х | X | X | X | X | X | X | Х | Use Days 2-8 |
| Subject | Χ | X | | | | X | | X | X | Use Days 2, 6, and 8 |
| Subject | X | X | | | X | | | | | Do Not Use |
| Subject | Χ | | | Χ | | Χ | | | Χ | Do Not Use |

 Table 2.2
 Examples of Visit 2 Day Selection for Activity Monitor Analysis

| Days With Valid Activity Monitoring Data | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Day of Activity | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | Use/Do Not Use |
| Monitoring | | | | | | | | | | |
| Target Study | Visit 2 | Study Day | Study Day | Study Day 4 | Study Day | Study | Study | Study | Study | |
| Day | | 2 | 3 | | 5 | Day 6 | Day 7 | Day 8 | Day 9 | |
| Subject <b>PP</b> | Χ | X | X | X | X | Χ | Χ | Χ | Χ | Use Days 2-8 |
| Subject | Χ | | | X | X | Χ | Χ | | | Use Days 4-8 |
| Subject | | X | X | X | X | Χ | Χ | Χ | Χ | Use Days 2-8 |
| Subject | Χ | X | | | | Χ | | Χ | X | Use Days 2, 6, |
| | | | | | | | | | | and 8 |
| Subject | Χ | X | | | X | | | | | Do Not Use |
| Subject | Χ | | | X | | Χ | | | Χ | Do Not Use |

 Table 2.3
 Examples of Visit 3 Day Selection for Activity Monitor Analysis

| Days With Valid Activity Monitoring Data | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Day of Activity | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | Use/Do Not Use |
| Monitoring | | | | | | | | | | |
| Target Study | Visit 3 | Study Day | Study Day | Study Day | Study Day | Study | Study | Study | Study | |
| Day | | 29 | 30 | 31 | 32 | Day 33 | Day 34 | Day 35 | Day 36 | |
| Subject <b>P</b> | Χ | Χ | Χ | X | Χ | Χ | Χ | Χ | X | Use Days 2-8 |
| Subject | Χ | | | X | Χ | Χ | Χ | | | Use Days 4-8 |
| Subject | | Χ | X | X | X | Χ | Χ | Χ | Χ | Use Days 2-8 |
| Subject | Χ | Χ | | | | Χ | | Χ | Χ | Use Days 2, 6, |
| | | | | | | | | | | and 8 |
| Subject | Χ | X | | | Χ | | | | | Do Not Use |
| Subject | Χ | | | X | | Χ | | | Χ | Do Not Use |

 Table 2.4
 Examples of Visit 5 Day Selection for Activity Monitor Analysis

| | | | D | ays With Valid | d Activity Mor | nitoring Dat | a | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Day of Activity | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | Use/Do Not Use |
| Monitoring | | | | | | | | | | |
| Target Study | Study | Study Day | Study Day | Study Day | Study Day | Study | Study | Study Day | Visit 5 | |
| Day | Day | 161 | 162 | 163 | 164 | Day 165 | Day 166 | 167 | | |
| _ | 160 | | | | | | | | | |
| Subject PP | Χ | Χ | X | X | Χ | Χ | X | Χ | Χ | Use Days 2-8 |
| Subject | Χ | | | X | X | Χ | Χ | | | Use Days 4-8 |
| Subject | | Χ | X | X | X | Χ | Χ | Χ | Χ | Use Days 2-8 |
| Subject | Χ | X | | | | Χ | | Χ | Χ | Use Days 2, 6, |
| | | | | | | | | | | and 8 |
| Subject | Χ | Χ | | | X | | | | | Do Not Use |
| Subject | Χ | | | Χ | | Χ | | | X | Do Not Use |

# 10.5.4. Safety

# **Adverse Events**

# **AE's OF Special Interest**

 AE groups of special interest have been defined as AEs which have specified areas of interest for UMEC or VI or the overall COPD population. Groups which are not SMQs are made up of a selection of preferred terms (PTs) defined by GSK. The complete list, including the preferred terms which contribute to each of the groups will be provided by Global Clinical Safety and Pharmacovigilance (GCSP) using the MedDRA version at the time of reporting. This will be finalised prior to unblinding.

| Special Interest AE<br>Group | Subgroup | Sub-SMQ | SMQ Group |
|---|---|---|---|
| Anticholinergic syndrome | | | Anticholinergic syndrome (SMQ) |
| Asthma/bronchospasm | | | Asthma/bronchospasm (SMQ) |
| Paradoxical bronchospasm | | | |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Arrhythmia<br>related<br>investigations,<br>signs and<br>symptoms<br>(SMQ) | Arrhythmia related investigations, signs and symptoms (SMQ) |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Bradyarrhythmia<br>terms,<br>nonspecific<br>(SMQ) | Bradyarrhythmia terms,<br>nonspecific (SMQ) |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Conduction defects (SMQ) | Conduction defects (SMQ) |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Disorders of sinus node function (SMQ) | Disorders of sinus node function (SMQ) |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Cardiac<br>arrhythmia<br>terms,<br>nonspecific<br>(SMQ) | Cardiac arrhythmia terms,<br>nonspecific (SMQ) |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Supraventricular tachyarrhythmias (SMQ) | Supraventricular tachyarrhythmias (SMQ) |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Tachyarrhythmia terms, | Tachyarrhythmia terms, nonspecific (SMQ) |

| Special Interest AE<br>Group | Subgroup | Sub-SMQ | SMQ Group |
|---|---|---|---|
| | | nonspecific<br>(SMQ) | |
| Cardiovascular effects | Cardiac<br>Arrhythmia | Ventricular<br>tachyarrhythmias<br>(SMQ) | Ventricular tachyarrhythmias<br>(SMQ) |
| Cardiovascular effects | Cardiac Failure | | Cardiac failure (SMQ) |
| Cardiovascular effects | Cardiac<br>Ischaemia | | Ischaemic heart disease (SMQ) |
| Cardiovascular effects | Hypertension | | Hypertension (SMQ) |
| Cardiovascular effects | Stroke | | Central nervous system haemorrhages and cerebrovascular conditions (SMQ) |
| Pneumonia | | | Infective pneumonia (SMQ) |
| LRTI excluding infective pneumonia | | | |
| Ocular effects (antimuscarinic) | | | Glaucoma (SMQ) |
| Effects on glucose | | | Hyperglycaemia/new onset diabetes mellitus (SMQ) |
| Effects on potassium | | | |
| Gastrointestinal obstruction | | | Gastrointestinal obstruction (SMQ) |
| Hypersensitivity | | | |
| Tremor | | | |
| Urinary retention | | | |

# Exposure

#### **Exposure Duration**

• Number of days of exposure to study drug will be calculated based on the formula:

Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- If a subject's overall exposure stop date is missing it will be assumed to be the latest recorded exposure start or stop date in the database.
- If a subject's overall exposure start date is missing then it will be assumed to be their Day 1 visit date (Visit 2).
- If a subject received a treatment other than the randomized treatment during the study, the exposure will still be calculated based on overall exposure start and stop dates.
- If the dose counter start=dose counter stop then it will be assumed that no doses were taken from that container.

# **Exposure Categories**

The following exposure categories will be derived:

1-84 days, 85-168 days, >168 days

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as receiving treatment at the final on-treatment clinic visit (Visit 5) and completion of the follow-up contact (Visit 6).</li> <li>Withdrawn subjects will not be replaced in the study.</li> </ul> |
| | <ul> <li>With the exception of the responder analyses, the minimum data required will be a baseline evaluation and at least one post-baseline evaluation. Note that this is not the case for the responder definition, see Section 10.6.2.3 for details.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays unless all data for a specific visit are missing in which case the visit is not displayed in the listing.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> <li>No imputation will be made for any missing numerical data. Missing data will generally not be considered in the calculation of percentages (i.e., the denominator will not include subjects who have missing data at a given time point).</li> </ul> </li> </ul> |

# 10.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | stop date of study treatment; in this case the study treatment stop date will be used. • Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

# 10.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.6.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Responder | <ul> <li>Subjects with a missing baseline will have responder status as missing</li> <li>Subjects with missing post-baseline data at a time point and a subsequent non-missing assessment will not be considered a responder or non-responder but will be left as missing at that time point</li> </ul> |
| | <ul> <li>Subjects with a missing post-baseline assessment with no subsequent non-missing assessments will be considered a non-responder for that and all subsequent time points.</li> <li>Subjects with a baseline but all missing post-baseline data will be</li> </ul> |
| | considered a non-responder at all time points. |

# 10.7. Appendix 7: Abbreviations & Trade Marks

# 10.7.1. Abbreviations

| Abbreviation | Description |
|------------------|--------------------------------------------------------|
| A&R | Analysis and Reporting |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ANCOVA | Analysis of Covariance |
| ASE | All Subjects Enrolled |
| ATC | Anatomical-Therapeutic-Chemical |
| BDI | Baseline Dyspnea Index |
| CAT | COPD Assessment Test |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| COPD | Chronic Obstructive Pulmonary Disease |
| CSR | Clinical Study Report |
| CV | Cardiovascular |
| DBF | Database Freeze |
| DM | Data Management |
| DPI | Dry Powder Inhaler |
| eCRF | Electronic Case Record Form |
| EXACT | Exacerbations of Chronic Pulmonary Disease Tool |
| FEV <sub>1</sub> | Forced Expiratory Volume in One Second |
| FVC | Forced Vital Capacity |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GOLD | Global Initiative for Chronic Obstructive Lung Disease |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| IA | Interim Analysis |
| ICS | Inhaled Corticosteroid |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| KR | Kenwood Roger |
| LRTI | Lower Respiratory Tract Infection |
| LS | Least-square |
| mcg | Microgram |
| MMRM | Mixed Model Repeated Measures |
| PD | Protocol Deviation |
| PDMP | Protocol Deviation Management Plan |
| PRO | Patient Reported Outcomes |
| QD | Once Daily |
| QoL | Quality of Life |

| Abbreviation | Description |
|--------------|--------------------------------------------|
| RAMOS | Randomization & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| RMC | Respiratory Medication Classification |
| RTF | Rich Text Format |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SAL | Salmeterol |
| SDL | Source Data Lock |
| SDTM | Study Data Tabulation Model |
| SE | Standard Error |
| SGRQ | St. George Respiratory Questionnaire |
| SGRQ-C | SGRQ for COPD patients |
| SI | System Independent |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| TDI | Transition Dyspnea Index |
| TFL | Tables, Figures & Listings |
| UMEC | Umeclidinium Bromide (GSK573719) |
| VI | Vilanterol Trifenatate |

# 10.7.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| DISKUS |
| ELLIPTA |

Trademarks not owned by the GlaxoSmithKline Group of Companies
SAS

# 10.8. Appendix 8: List of Data Displays

# 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-----------------------|------------|
| Study Population | 1.1 to 1.n 1.1 to 1.n | |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n 3.1 to 3.n | |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

# 10.8.2. Deliverables

| Delivery | Description |
|----------|--------------------------------------|
| SAC | Final Statistical Analysis Complete. |

# 10.8.3. Study Population Tables

| Study P | opulation T | ables | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| Subject | Subject Disposition | | | |
| 1.1 | ASE | Summary of Study Populations | | SAC |
| 1.2 | ASE | Summary of Screen Failures and Run-in failures | | SAC |
| 1.3 | ITT | Summary of Attendance/Telephone Contact at Each Visit | | SAC |
| 1.4 | ITT | Summary of Completion and Premature Discontinuation of Study Treatment | | SAC |
| 1.5 | ITT | Summary of Study Completion and Withdrawal | | SAC |
| 1.6 | ITT | Summary of Number of Subjects by Geographical Region, Country and Center | | SAC |
| 1.7 | ASE | Summary of Inclusion/ Exclusion/ Randomization Criteria Deviations for Screen or Run-<br>in failures | | SAC |
| 1.8 | ITT | Summary of Inclusion/ Exclusion/ Randomization Criteria Deviations | | SAC |
| 1.9 | ITT | Summary of Important Protocol Deviations | | SAC |
| Demogra | aphy | | 1 | |
| 1.10 | ITT | Summary of Demographic Characteristics | | SAC |
| 1.11 | ITT | Summary of Race and Racial Combinations | | SAC |
| 1.12 | ITT | Summary of Race and Racial Combination Details | | SAC |
| Medical | Condition & | & Concomitant Medications | | |
| 1.13 | ITT | Summary of Current Medical Conditions | | SAC |
| 1.14 | ITT | Summary of Past Medical Conditions | | SAC |
| 1.15 | ITT | Summary of Cardiovascular Risk Factors | | SAC |
| 1.16 | ITT | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| 1.17 | ITT | Summary of COPD History at Screening | Include Duration of COPD and COPD type | SAC |
| 1.18 | ITT | Summary of COPD Exacerbation History at Screening | 71 | SAC |

| Study P | opulation T | ables | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| 1.19 | ITT | Summary of Smoking Status and History at Screening | | SAC |
| 1.20 | ITT | Summary of Long-acting Bronchodilator Usage during the Run-in (Randomization Strata) | | |
| 1.21 | ITT | Summary of Concomitant Medications Not Given for a COPD Exacerbation Taken Pre-<br>Treatment | | SAC |
| 1.22 | ITT | Summary of Concomitant Medications Not Given for a COPD Exacerbation Taken Ontreatment | | SAC |
| 1.23 | ITT | Summary of Concomitant Medications Not Given for a COPD Exacerbation Taken Post-treatment | | |
| 1.24 | ITT | Summary of Concomitant Medications Given for a COPD Exacerbation Taken Pretreatment | | SAC |
| 1.25 | ITT | Summary of Concomitant Medications Given for a COPD Exacerbation Taken Ontreatment | | SAC |
| 1.26 | ITT | Summary of Concomitant Medications Given for a COPD Exacerbation Taken Post-treatment | | SAC |
| Baseline | Severity | | | |
| 1.27 | ITT | Summary of Screening Lung Function Test Results | | SAC |
| 1.28 | ITT | Summary of GOLD Grade 1-4, GOLD CAT Category A-D and Reversibility at Screening | | SAC |
| 1.29 | ITT | Summary of GOLD Grade 1-4, GOLD CAT Category A-D and Reversibility at Screening by Country | | SAC |
| 1.30 | ITT | Summary of CAT Score at Screening | | SAC |
| Complia | ınce | | | |
| 1.31 | ITT | Summary of Device and Overall Percentage Treatment Compliance | | SAC |

# 10.8.4. Efficacy Tables

| Efficac | cy: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| | 1 | <u></u> | | |
| 2.01 | ITT | Summary of Baseline FEV1 (L) | | SAC |
| 2.02 | ITT | Summary of Trough FEV1 (L) | | SAC |
| 2.03 | ITT | Analysis of Trough FEV1 (L) | | SAC |
| 2.04 | ITT | Covariance Parameter Estimates for Repeated Measures Analysis of Trough FEV1 (L) | | SAC |
| 2.05 | ITT | Type III Tests of Fixed Effects for Repeated Measures Analysis of Trough FEV1 (L) | | SAC |
| 2.06 | ITT | Significance Levels for Interactions of Treatment with Baseline FEV1, Geographical Region and Stratum for Trough FEV1 (L) | | SAC |
| 2.07 | ITT | Analysis of Ratio (Trough FEV1/Baseline FEV1) | | SAC |
| 2.08 | ITT | Summary of Baseline FVC (L) | | SAC |
| 2.09 | ITT | Summary of Trough FVC (L) | | SAC |
| 2.10 | ITT | Analysis of Trough FVC (L) | | SAC |
| 2.11 | ITT | Summary of Baseline IC (L) | | SAC |
| 2.12 | ITT | Summary of Trough IC (L) | | SAC |
| 2.13 | ITT | Analysis of Trough IC (L) | | SAC |
| BDI/TE | DI | | | |
| 2.14 | ITT | Summary of BDI Focal Score | | SAC |
| 2.15 | ITT | Summary of TDI Focal Score | | SAC |
| 2.16 | ITT | Analysis of TDI Focal Score | | SAC |
| 2.17 | ITT | Summary and Analysis of Proportion of Responders According to TDI Focal Score | | SAC |
| E-RS | | | | |
| 2.18 | ITT | Summary of Four-Weekly Mean E-RS Total Score | | SAC |
| 2.19 | ITT | Summary of Four-Weekly Mean E-RS Breathlessness Score | | SAC |

| Efficac | Efficacy: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| 2.20 | ITT | Summary of Four-Weekly Mean E-RS Cough and Sputum Score | | SAC |
| 2.21 | ITT | Summary of Four-Weekly Mean E-RS Chest Score | | SAC |
| 2.22 | ITT | Analysis of Four-Weekly Mean E-RS Total Score | | SAC |
| 2.23 | ITT | Analysis of Four-Weekly Mean E-RS Breathlessness Score | | SAC |
| 2.24 | ITT | Analysis of Four-Weekly Mean E-RS Cough and Sputum Score | | SAC |
| 2.25 | ITT | Analysis of Four-Weekly Mean E-RS Chest Score | | SAC |
| 2.26 | ITT | Summary and Analysis of Proportion of Responders According To E-RS Total Score | | SAC |
| 2.27 | ITT | Summary and Analysis of Proportion of Responders According To E-RS Breathlessness Score | | SAC |
| 2.28 | ITT | Summary and Analysis of Proportion of Responders According To E-RS Cough and Sputum Score | | SAC |
| 2.29 | ITT | Summary and Analysis of Proportion of Responders According To E-RS Chest Score | | SAC |
| SGRQ | -C | | | |
| 2.30 | ITT | Summary of Baseline SGRQ Scores | | SAC |
| 2.31 | ITT | Summary of SGRQ Total Score | | SAC |
| 2.32 | ITT | Summary of SGRQ Symptoms Score | | SAC |
| 2.33 | ITT | Summary of SGRQ Activity Score | | SAC |
| 2.34 | ITT | Summary of SGRQ Impacts Score | | SAC |
| 2.35 | ITT | Analysis of SGRQ Total Score | | SAC |
| 2.36 | ITT | Summary and Analysis of Proportion of Responders According To SGRQ Total Score | | SAC |
| CAT | | | | |
| 2.37 | ITT | Summary of CAT Score | Include Baseline | SAC |
| 2.38 | ITT | Analysis of CAT Score | | SAC |
| 2.39 | ITT | Summary and Analysis of Proportion of Responders According To CAT Score | | SAC |

| Efficacy: Tables | | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| COPD | COPD Exacerbations | | | |
| 2.40 | ITT | Summary of On-Treatment COPD Exacerbations | | SAC |
| 2.41 | ITT | Summary of Post-Treatment COPD Exacerbations | | SAC |
| 2.42 | ITT | Summary and Analysis of Time to First On-Treatment Mild/Moderate/Severe COPD Exacerbation | | SAC |
| 2.43 | ITT | Summary and Analysis of Time to First On-Treatment Moderate/Severe COPD Exacerbation | | SAC |
| 2.44 | ITT | Summary and Analysis of Time to First On-Treatment Severe COPD Exacerbation | | SAC |
| 2.45 | ITT | Annual rate of on-treatment mild/moderate/severe exacerbations | | SAC |
| 2.46 | ITT | Annual rate of on-treatment moderate/severe exacerbations | | SAC |
| CID | | | | |
| 2.47 | ITT | Summary of Deterioration and Individual Components | Include all composites | SAC |
| 2.48 | ITT | Summary and Analysis of Time to First Decrease from Baseline of >=100ml in Trough FEV1 | | SAC |
| 2.49 | ITT | Summary and Analysis of Time to First Increase from Baseline of >=4 units in SGRQ Total Score | | SAC |
| 2.50 | ITT | Summary and Analysis of Time to First Increase from Baseline of >=2 units in CAT Score | | SAC |
| 2.51 | ITT | Summary and Analysis of Time to First Decrease of >=1 units in TDI | | SAC |
| 2.52 | ITT | Summary and Analysis of Time to First Deterioration (SGRQ, FEV1, EXAC (mod/sev)) | | SAC |
| 2.53 | ITT | Summary and Analysis of Time to First Deterioration (CAT, FEV1, EXAC (mod/sev)) | | SAC |
| 2.54 | ITT | Summary and Analysis of Time to First Deterioration (CAT, SGRQ, TDI, EXAC (mod/sev)) | | SAC |
| 2.55 | ITT | Summary of Deterioration Status at Day 30 | | SAC |
| 2.56 | ITT | Analysis of Four-Weekly Mean E-RS Total Score by Day 30 Deterioration Status | | SAC |

| Efficac | Efficacy: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| 2.57 | ITT | Analysis of Mean Number of Inhalations of Rescue use per Day using e-Diary Day 30 Deterioration Status | | SAC |
| 2.58 | ITT | Summary and Analysis of Time to First On-Treatment Moderate/Severe Exacerbation leading to hospitalisation by Day 30 Deterioration Status | | SAC |
| 2.59 | ITT | Summary and Analysis of Time to Mortality by Day 30 Deterioration Status | | SAC |
| Rescu | e Use | | | |
| 2.60 | ITT | Summary of Mean Number of Inhalations of Rescue Medication per Day using e-Diary | | SAC |
| 2.61 | ITT | Analysis of Mean Number of Inhalations of Rescue Medication per Day over Weeks 1-24 using e-Diary | | SAC |
| 2.62 | ITT | Summary of Percentage of Rescue-Free Days using e-Diary | | SAC |
| 2.63 | ITT | Analysis of Percentage of Rescue-Free Days over Weeks 1-24 using e-Diary | | SAC |
| 2.64 | ITT | Summary of Mean Number of Occurrences of Rescue Medication per Day using eMDI. | | SAC |
| 2.65 | ITT | Analysis of Mean Number of Occurrences of Rescue Medication per Day over Weeks 1-24 using eMDI | | SAC |
| 2.66 | ITT | Summary of Percentage of Rescue-Free Days using eMDI | | SAC |
| 2.67 | ITT | Analysis of Percentage of Rescue-Free Days over Weeks 1-24 using eMDI | | SAC |
| Subjec | t Global Ratir | ngs | | |
| 2.68 | ITT | Summary of Subject Global Rating of COPD Severity | | SAC |
| 2.69 | ITT | Summary and Analysis of Subject Global Rating of Change in COPD Severity | Use<br>gsk2834425/ctt116853<br>as reference | SAC |
| Physic | Physical Activity Monitor | | | |
| 2.70 | AM | Summary of Weekly Mean Step Count | | SAC |

| Efficac | Efficacy: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| 2.71 | AM | Analysis of Weekly Mean Step Count | | SAC |
| 2.72 | AM | Summary of Weekly Mean Duration of Light Physical Activity (Hours) | | SAC |
| 2.73 | AM | Analysis of Weekly Mean Duration of Light Physical Activity (Hours) | | SAC |
| 2.74 | AM | Summary of Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) | | SAC |
| 2.75 | AM | Analysis of Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) | | SAC |
| 2.76 | AM | Summary of Weekly Mean Total Energy Expenditure (kCal) | | SAC |
| 2.77 | AM | Analysis of Weekly Mean Total Energy Expenditure (kCal) | | SAC |

# 10.8.5. Efficacy Figures

| Efficacy | Efficacy: Figures | | | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| Spirome | etry | | | |
| 2.01 | ITT | Box Plot of Change from Baseline in Trough FEV1 (L) at Week 24 | | SAC |
| 2.02 | ITT | Empirical Distribution Function Plot of Change from Baseline in Trough FEV1 (L) at Week 24 | | SAC |
| 2.03 | ITT | Least Squares Mean (95% CI) Change from Baseline in Trough FEV1 (L) | | SAC |
| 2.04 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Trough FEV1 (L) | | SAC |
| 2.05 | ITT | Least Squares Mean (95% CI) Change from Baseline in Trough FVC (L) | | SAC |
| 2.06 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Trough FVC (L) | | SAC |
| 2.07 | ITT | Least Squares Mean Change from Baseline (95% CI) in Trough IC (L) | | SAC |

| Efficacy | : Figures | | | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| 2.08 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Trough IC (L) | | SAC |
| BDI/TDI | | | | |
| 2.09 | ITT | Least Squares Means (95% CI) TDI Focal Score | | SAC |
| 2.10 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in TDI Focal Score | | SAC |
| E-RS | | | | |
| 2.11 | ITT | Least Squares Mean Change from Baseline (95% CI) in Four-Weekly Mean E-RS Total Score | | SAC |
| 2.12 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Four-Weekly Mean E-RS Total Score | | SAC |
| 2.13 | ITT | Least Squares Mean Change from Baseline (95% CI) in Four-Weekly Mean E-RS Breathlessness Score | | SAC |
| 2.14 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Four-Weekly Mean E-RS Breathlessness Score | | SAC |
| 2.15 | ITT | Least Squares Mean Change from Baseline (95% CI) in Four-Weekly Mean E-RS Cough and Sputum Score | | SAC |
| 2.16 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline ) in Four-Weekly Mean E-RS Cough and Sputum Score | | SAC |
| 2.17 | ITT | Least Squares Mean Change from Baseline (95% CI) in Four-Weekly Mean E-RS Chest Score | | SAC |
| 2.18 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Four-Weekly Mean E-RS Chest Score | | SAC |
| SGRQ | | | | |
| 2.19 | ITT | Least Squares Mean (95% CI) Change from Baseline in SGRQ Total Score | | SAC |
| 2.20 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in SGRQ Total Score | | SAC |
| | : Figures Popu- lation | Title | Programming<br>Note | Deliverable |
|---|---|---|---|---|
| CAT | | | | |
| 2.21 | ITT | Least Squares Mean Change from Baseline (95% CI) in CAT Score | | SAC |
| 2.22 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline ) in CAT Score | | SAC |
| COPD E | xacerbation | S | | |
| 2.23 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Mild/Moderate/Severe COPD Exacerbation (Days) | | SAC |
| 2.24 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Moderate/Severe COPD Exacerbation (Days) | | SAC |
| 2.25 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Severe COPD Exacerbation (Days) | | SAC |
| CID | | | | |
| 2.26 | ITT | Kaplan-Meier Plot of Time to First Decrease from Baseline of >=100ml in Trough FEV1 | | SAC |
| 2.27 | ITT | Kaplan-Meier Plot of Time to First Increase from Baseline of >=4 units in SGRQ Total Score | | SAC |
| 2.28 | ITT | Kaplan-Meier Plot of Time to First Increase from Baseline of >=2 units in CAT Score | | SAC |
| 2.29 | ITT | Kaplan-Meier Plot of Time to First Decrease of >=1 units in TDI | | SAC |
| 2.30 | ITT | Kaplan-Meier Plot of Time to First Deterioration (SGRQ, FEV1, EXAC (mod/sev)) (Days) | | SAC |
| 2.31 | ITT | Kaplan-Meier Plot of Time to First Deterioration (CAT, FEV1, EXAC (mod/sev)) (Days) | | SAC |
| 2.32 | ITT | Kaplan-Meier Plot of Time to First Deterioration (CAT, SGRQ, TDI, EXAC (mod/sev)) (Days) | | SAC |
| 2.33 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Moderate/Severe Exacerbation Leading to Hospitalisation by Day 30 Deterioration Status | | SAC |
| 2.35 | ITT | Kaplan-Meier Plot of Time to Mortality by Day 30 Deterioration Status | | SAC |
| Rescue | Use | | | |
| 2.36 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Mean Number of Inhalations of Rescue Medication per Day over Weeks 1-24 using e-Diary | | SAC |

| Efficacy | : Figures | | | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| 2.37 | ITT | Least Squares Mean (95% CI) Change from Baseline in Percentage of Rescue-Free Days over Weeks 1-24 using e-Diary | | SAC |
| 2.38 | ITT | Least Squares Mean (95% CI) Treatment Difference in Change from Baseline in Mean Number of Occurrences of Rescue Medication per Day over Weeks 1-24 using eMDI | | SAC |
| 2.39 | ITT | Least Squares Mean (95% CI) Change from Baseline in Percentage of Rescue-Free Days over Weeks 1-24 using eMDI | | SAC |
| Physica | I Activity Mo | nitor | | |
| 2.40 | ITT | Histograms of Change from Baseline in Weekly Mean Step Count at Week 1, Week 4 and Week 24 by Treatment Group | | SAC |
| 2.41 | ITT | Histograms of Change from Baseline in Weekly Mean Duration of Light Physical Activity (Hours) at Week 1, Week 4 and Week 24 by Treatment Group | | SAC |
| 2.42 | ITT | Histograms of Change from Baseline in Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) at Week 1, Week 4 and Week 24 by Treatment Group | | SAC |
| 2.43 | ITT | Histograms of Change from Baseline in Weekly Mean Total Energy Expenditure (kCal) at Week 1, Week 4 and Week 24 by Treatment Group | | SAC |
| 2.44 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Step Count | | SAC |
| 2.45 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Duration of Light Physical Activity (Hours) | | SAC |
| 2.46 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) | | SAC |
| 2.47 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Total Energy Expenditure (kCal) | | SAC |

# 10.8.6. Safety Tables

| Safety Table | es | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| Exposure | | | | |
| 3.01 | ITT | Summary of Exposure | | SAC |
| Adverse Ev | ents | | | |
| 3.02 | ITT | Overview of Adverse Events | | SAC |
| 3.03 | ITT | Summary of On-treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.04 | ITT | Summary of Post-treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.05 | ITT | Summary of On-treatment Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.06 | ITT | Summary of Pre-treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.07 | ITT | Summary of On-treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.08 | ITT | Summary of On-treatment Fatal Serious Adverse Events by System Organ Class and Preferred Term | | SAC |

| No. | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
|---|---|---|---|---|
| 3.09 | ITT | Summary of On-treatment Serious Adverse Events (Serious, Drug-Related Serious and Fatal) by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 3.10 | ASE | Summary of Pre-treatment Adverse Events Leading Withdrawal from the Study by System Organ Class and Preferred Term | | SAC |
| 3.11 | ITT | Summary of On-treatment Drug-related Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.12 | ITT | Summary of On-treatment Drug-related Fatal Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.13 | ITT | Summary of On-treatment Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from the Study by System Organ Class and Preferred Term | | SAC |
| 3.14 | ITT | Summary of On-treatment Adverse Events of Special Interest | | SAC |
| 3.15 | ITT | Summary of On-treatment Serious Adverse Events of Special Interest | | SAC |
| 3.16 | ASE | Relationship between Adverse Event System Organ Class, Preferred Term and Verbatim Text | | SAC |
| 3.17 | ITT | Summary of Common (>=3%) On-treatment Non-Serious Drug-related Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |

| Safety Table | Safety Tables | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| 3.18 | ITT | Summary of Common (>=3%) On-treatment Serious Adverse Events by Overall Frequency | | SAC |
| 3.19 | ITT | Summary of Common (>=3%) On-treatment Serious Drug-related Adverse Events by Overall Frequency | | SAC |
| 3.20 | ITT | Summary of the 10 Most Frequent On-treatment Adverse Events in Each Treatment Group | | SAC |
| 3.21 | ITT | Summary of On-treatment Adverse Events by System Organ Class, Preferred Term and Age Subgroup | | SAC |
| 3.22 | ITT | Summary of On-treatment Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | SAC |
| 3.33 | ITT | Summary of On-treatment Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | SAC |

## 10.8.7. Safety Figures

| Safety: F | Safety: Figures | | | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| 3.01 | ITT | Adverse Event Incidence Rates and Relative Risks | | SAC |

## 10.8.8. ICH Listings

| ICH : L | _istings | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| Study | Population | on | | |
| 1. | ITT | Listing of Subjects who Discontinued Study Treatment | | SAC |
| 2. | ITT | Listing of Reasons for Withdrawal | | SAC |
| 3. | ASE | Listings of Reasons for Withdrawal – Subjects Randomised but not in the Intent-to-Treat Population | | SAC |
| 4. | ITT | Listing of the Follow-up Contact | | SAC |
| 5. | ITT | Listing of Important Protocol Deviations | | SAC |
| 6. | ITT | Listing of Subjects with Inclusion, Exclusion or Randomisation Criteria Deviations | | SAC |
| 7. | ITT | Listing of Subjects for whom the Treatment Blind was Broken | | SAC |
| 8. | ITT | Listing of Randomised and Actual Treatments | | SAC |
| 9. | ITT | Listing of Overall Treatment Compliance | | SAC |
| 10. | ITT | Listing of Demographic Characteristics | | SAC |
| 11. | ITT | Listing of Race | | SAC |
| 12. | ITT | Listing of Medical Conditions | | SAC |

| ICH : L | istings | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| 13. | ITT | Listing of Cardiovascular Risk Factors | | SAC |
| 14. | ITT | Listing of Family History of Cardiovascular Risk Factors | | SAC |
| 15. | ITT | Listing of Concomitant Medications Given for a COPD Exacerbation | | SAC |
| 16. | ITT | Listing of Concomitant Medications Not Given for a COPD Exacerbation | | SAC |
| 17. | ITT | Relationship between ATC Level 1, ingredient and verbatim text Non-COPD medications | | SAC |
| 18. | ITT | Listing of COPD History | Include COPD duration and COPD type | SAC |
| 19. | ITT | Listing of Smoking History and Smoking Status | | SAC |
| Study | Population | on | | |
| 20. | ITT | Listing of Screening Lung Function Test Results | | SAC |
| 21. | ITT | Listing of GOLD Grade/Categories, Reversibility and long-acting bronchodilator usage stratum at Screening | | SAC |
| 22. | ITT | Listing of Derived FEV1 (L) Endpoints | | SAC |
| 23. | ITT | Listing of Derived FVC (L) Endpoints | | SAC |
| 24. | ITT | Listing of Derived IC (L) Endpoints | | SAC |

| ICH : L | istings | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| 25. | ITT | Listing of Derived Rescue Use Endpoints (eDiary) | | SAC |
| 26. | ITT | Listing of Derived Rescue Use Endpoints (eMDI) | | SAC |
| 27. | ITT | Listing of Derived E-RS Scores | | SAC |
| 28. | ITT | Listing of CAT Scores | Include Screening | SAC |
| 29. | ITT | Listing of SGRQ Scores | | SAC |
| 30. | ITT | Listing of TDI Scores | | SAC |
| Expos | ure | | | |
| 31. | ITT | Listing of Exposure | | SAC |
| Adver | se Events | S | | |
| 32. | ITT | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 33. | ITT | Listing of All Adverse Events | | SAC |
| 34. | ITT | Listing of Non-fatal Serious Adverse Events | | SAC |
| 35. | ITT | Listing of Fatal Serious Adverse Events | | SAC |
| 36. | ITT | Listing of Adverse Events Leading to Discontinuation of Study Treatment or Withdrawal from the Study | | SAC |

| ICH : I | istings | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| 37. | ITT | Listing of On-treatment Drug-Related Adverse Events | | SAC |
| 38. | ITT | Listing of Reasons for Considering as a Serious Adverse Event | | |
| Inhale | r Malfund | ctions | 1 | |
| 39. | ITT | Listing of Potential DPI Inhaler Malfunctions | | SAC |
| COPD | Exacerb | ations | | |
| 40. | ITT | Listing of COPD Exacerbations | | SAC |
| Pneun | nonia and | d Chest X-ray | | |
| 41. | ITT | Listing of Chest X-ray Data | | SAC |
| 42. | ITT | Listing of All Pneumonia Data | | SAC |
| Liver I | Events: N | lote only produced if there is a Liver Event | | |
| 43. | ITT | Listing of Liver Events | | SAC |
| 44. | ITT | Listing of Liver Event Information for RUCAM Score | | SAC |
| 45. | ITT | Listing of Liver Biopsy | | SAC |
| 46. | ITT | Listing of Liver Imaging Details | | SAC |
| | | <u>I</u> | | |

| ICH : Listings | | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| Cardiovascular Events: Note only produced if there is a Cardiovascular Event | | | | |
| 47. | ITT | Listing of Myocardial Infarction/Unstable Angina | Include under patient profiles in HARP | SAC |
| 48. | ITT | Listing of Congestive Heart Failure | Include under patient profiles in HARP | SAC |
| 49. | ITT | Listing of Arrhythmias | Include under patient profiles in HARP | SAC |
| 50. | ITT | Listing of Valvulopathy | Include under patient profiles in HARP | SAC |
| 51. | ITT | Listing of Pulmonary Hypertension | Include under patient profiles in HARP | SAC |
| 52. | ITT | Listing of Cerebrovascular Events/Stroke and Transient Ischemic Attack | Include under patient profiles in HARP | SAC |

| ICH : L | ICH : Listings | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| 53. | ITT | Listing of Peripheral Arterial Thromboembolism | Include under patient profiles in HARP | SAC |
| 54. | ITT | Listing of Deep Venous Thrombosis/Pulmonary Embolism | Include under patient profiles in HARP | SAC |
| 55. | ITT | Listing of Revascularisation | Include under patient profiles in HARP | SAC |
| 56. | ITT | Listing of All cause deaths | Include under patient profiles in HARP | SAC |

## 10.8.9. Non-ICH Listings

| Non-IC | H : Listing | ys . | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming<br>Note | Deliverable |
| Study | Study Population | | | |
| 57. | ITT | Listing of Treatment Misallocations | | SAC |
| 58. | ITT | Listing of Raw FEV1 (L) and FVC (L) Data | | SAC |
| 59. | ITT | Listing of Raw IC (L) Data | | SAC |
| 60. | ITT | Listing of Adverse Event of Special Interest Group, Subgroup, Sub-SMQ and Preferred Term | | SAC |
| 61. | AM | Listing of Physical Activity Monitoring Data | | SAC |

### 10.8.10. Maintenance Naive

## 10.8.1. Study Population Tables

| Study Po | Study Population Tables | | |
|---|---|---|---|
| No. | No. Population Title Programming Note | | |
| Subject D | Disposition | | |
| 1.33 | ITT | Summary of Study Completion and Withdrawal | SAC |

| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
|---|---|---|---|---|
| Demogra | aphy | · | <u> </u> | |
| 1.34 | ITT | Summary of Demographic Characteristics | | SAC |
| 1.35 | ITT | Summary of Maintenance Naive Status | | SAC |
| Medica | al Condition | & Concomitant Medications | | |
| 1.36 | ITT | Summary of Current Medical Conditions | | SAC |
| 1.37 | ITT | Summary of Cardiovascular Risk Factors | | SAC |
| 1.38 | ITT | Summary of COPD History at Screening | Include Duration of COPD and COPD type | SAC |
| 1.39 | ITT | Summary of COPD Exacerbation History at Screening | | SAC |
| 1.40 | ITT | Summary of Smoking Status and History at Screening | | SAC |
| Baseline | Severity | | <u> </u> | |
| 1.41 | ITT | Summary of Screening Lung Function Test Results | | SAC |
| 1.42 | ITT | Summary of GOLD Grade 1-4, GOLD CAT Category A-D and Reversibility at Screening | | SAC |
| 1.43 | ITT | Summary of CAT Score at Screening | | SAC |
| Compliar | nce | 1 | | |
| 1.44 | ITT | Summary of Device and Overall Percentage Treatment Compliance | | SAC |

# 10.8.2. Efficacy Tables

| Efficacy: Tables | | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| 2.78 | ITT | Summary of Baseline FEV1 (L) | | SAC |
| 2.79 | ITT | Summary of Trough FEV1 (L) | | SAC |
| 2.80 | ITT | Analysis of Trough FEV1 (L) | | SAC |
| 2.81 | ITT | Analysis of Ratio (Trough FEV1/Baseline FEV1) | | SAC |
| 2.82 | ITT | Summary of Baseline FVC (L) | | SAC |
| 2.83 | ITT | Summary of Trough FVC (L) | | SAC |
| 2.84 | ITT | Analysis of Trough FVC (L) | | SAC |
| 2.85 | ITT | Summary of Baseline IC (L) | | SAC |
| 2.86 | ITT | Summary of Trough IC (L) | | SAC |
| 2.87 | ITT | Analysis of Trough IC (L) | | SAC |
| BDI/TDI | | | · | |
| 2.88 | ITT | Summary of BDI Focal Score | | SAC |
| 2.89 | ITT | Summary of TDI Focal Score | | SAC |

| Efficacy: | lables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| 2.90 | ITT | Analysis of TDI Focal Score | | SAC |
| 2.91 | ITT | Summary and Analysis of Proportion of Responders According to TDI Focal Score | | SAC |
| E-RS | | | | |
| 2.92 | ITT | Summary of Four-Weekly Mean E-RS Total Score | | SAC |
| 2.93 | ITT | Analysis of Four-Weekly Mean E-RS Total Score | | SAC |
| 2.94 | ITT | Summary and Analysis of Proportion of Responders According To E-RS Total Score | | SAC |
| SGRQ-C | | | | |
| 2.95 | ITT | Summary of Baseline SGRQ Scores | | SAC |
| 2.96 | ITT | Summary of SGRQ Total Score | | SAC |
| 2.97 | ITT | Analysis of SGRQ Total Score | | SAC |
| 2.98 | ITT | Summary and Analysis of Proportion of Responders According To SGRQ Total Score | | SAC |
| CAT | | | | |
| 2.99 | ITT | Summary of CAT Score | Include Baseline | SAC |
| 2.100 | ITT | Analysis of CAT Score | | SAC |

| Efficacy: | Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| 2.101 | ITT | Summary and Analysis of Proportion of Responders According To CAT Score | | SAC |
| COPD Ex | acerbations | | | |
| 2.102 | ITT | Summary of On-Treatment COPD Exacerbations | | SAC |
| 2.103 | ITT | Summary of Post-Treatment COPD Exacerbations | | SAC |
| 2.104 | ITT | Summary and Analysis of Time to First On-Treatment Mild/Moderate/Severe COPD Exacerbation | | SAC |
| 2.105 | ITT | Summary and Analysis of Time to First On-Treatment Moderate/Severe COPD Exacerbation | | SAC |
| 2.106 | ITT | Summary and Analysis of Time to First On-Treatment Severe COPD Exacerbation | | SAC |
| 2.107 | ITT | Annual rate of on-treatment moderate/severe exacerbations | | SAC |
| CID | | | | |
| 2.108 | ITT | Summary of Deterioration and Individual Components | Include all composites | SAC |
| 2.109 | ITT | Summary and Analysis of Time to First Decrease from Baseline of >=100ml in Trough FEV1 | | SAC |
| 2.110 | ITT | Summary and Analysis of Time to First Increase from Baseline of >=4 units in SGRQ Total Score | | SAC |
| 2.111 | ITT | Summary and Analysis of Time to First Increase from Baseline of >=2 units in CAT Score | | SAC |
| 2.112 | ITT | Summary and Analysis of Time to First Decrease of >=1 units in TDI | | SAC |

| Efficacy: | | | Programming Note | |
|---|---|---|---|---|
| No. | Population | Title | | Deliverable |
| 2.113 | ITT | Summary and Analysis of Time to First Deterioration (SGRQ, FEV1, EXAC (mod/sev)) | | SAC |
| 2.114 | ITT | Summary and Analysis of Time to First Deterioration (CAT, FEV1, EXAC (mod/sev)) | | SAC |
| 2.115 | ITT | Summary and Analysis of Time to First Deterioration (CAT, SGRQ, TDI, EXAC (mod/sev)) | | SAC |
| Rescue L | Jse | | | |
| 2.116 | ITT | Summary of Mean Number of Inhalations of Rescue Medication per Day using e-Diary | | SAC |
| 2.117 | ITT | Analysis of Mean Number of Inhalations of Rescue Medication per Day over Weeks 1-24 using e-Diary | | SAC |
| 2.118 | ITT | Summary of Percentage of Rescue-Free Days using e-Diary | | SAC |
| 2.119 | ITT | Analysis of Percentage of Rescue-Free Days over Weeks 1-24 using e-Diary | | SAC |
| 2.120 | ITT | Summary of Mean Number of Occurrences of Rescue Medication per Day using eMDI | | SAC |
| 2.121 | ITT | Analysis of Mean Number of Occurrences of Rescue Medication per Day over Weeks 1-24 using eMDI | | SAC |
| 2.122 | ITT | Summary of Percentage of Rescue-Free Days using eMDI | | SAC |
| 2.123 | ITT | Analysis of Percentage of Rescue-Free Days over Weeks 1-24 using eMDI | | SAC |

| Efficacy: | Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Note | Deliverable |
| Subject ( | Global Ratings | | | |
| 2.124 | ITT | Summary of Subject Global Rating of COPD Severity | | SAC |
| 2.125 | ITT | Summary and Analysis of Subject Global Rating of Change in COPD Severity | Use gsk2834425/ctt116853 as reference | SAC |
| Physical | Activity Monitor | | | |
| 2.126 | ITT | Summary of Weekly Mean Step Count | | SAC |
| 2.127 | ITT | Analysis of Weekly Mean Step Count | | SAC |
| 2.128 | ITT | Summary of Weekly Mean Duration of Light Physical Activity (Hours) | | SAC |
| 2.129 | ITT | Analysis of Weekly Mean Duration of Light Physical Activity (Hours) | | SAC |
| 2.130 | ITT | Summary of Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) | | SAC |
| 2.131 | ITT | Analysis of Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) | | SAC |
| 2.132 | ITT | Summary of Weekly Mean Total Energy Expenditure (kCal) | | SAC |
| 2.133 | ITT | Analysis of Weekly Mean Total Energy Expenditure (kCal) | | SAC |

# 10.8.3. Efficacy Figures

| Efficacy: | Figures | | | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming Note | Deliverable |
| Spiromet | ry | | | |
| 2.48 | ITT | Least Squares Mean (95% CI) Change from Baseline in Trough FEV1 (L) | | SAC |
| 2.49 | ITT | Least Squares Mean Change from Baseline (95% CI) in Trough FVC (L) | | SAC |
| 2.50 | ITT | Least Squares Mean Change from Baseline (95% CI) in Trough IC (L) | | SAC |
| BDI/TDI | | | | |
| 2.51 | ITT | Least Squares Means (95% CI) TDI Focal Score | | SAC |
| E-RS | | | | |
| 2.52 | ITT | Least Squares Mean Change from Baseline (95% CI) in Four-Weekly Mean E-RS Total Score | | SAC |
| SGRQ | | | | |
| 2.53 | ITT | Least Squares Mean (95% CI) Change from Baseline in SGRQ Total Score | | SAC |
| CAT | | | | |
| 2.54 | ITT | Least Squares Mean Change from Baseline (95% CI) in CAT Score | | SAC |
| COPD Ex | acerbations | | | |
| 2.55 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Mild/Moderate/Severe COPD Exacerbation (Days) | | SAC |
| 2.56 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Moderate/Severe COPD Exacerbation (Days) | | SAC |
| 2.57 | ITT | Kaplan-Meier Plot of Time to First On-Treatment Severe COPD Exacerbation (Days) | | SAC |

| Efficacy: | | | D | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming Note | Deliverable |
| CID | | | | |
| 2.58 | ITT | Kaplan-Meier Plot of Time to First Decrease from Baseline of >=100ml in Trough FEV1 | | SAC |
| 2.59 | ITT | Kaplan-Meier Plot of Time to First Increase from Baseline of >=4 units in SGRQ Total Score | | SAC |
| 2.60 | ITT | Kaplan-Meier Plot of Time to First Increase from Baseline of >=2 units in CAT Score | | SAC |
| 2.61 | ITT | Kaplan-Meier Plot of Time to First Decrease of >=1 units in TDI | | SAC |
| 2.62 | ITT | Kaplan-Meier Plot of Time to First Deterioration (SGRQ, FEV1, EXAC (mod/sev)) (Days) | | SAC |
| 2.63 | ITT | Kaplan-Meier Plot of Time to First Deterioration (CAT, FEV1, EXAC (mod/sev)) (Days) | | SAC |
| 2.64 | ITT | Kaplan-Meier Plot of Time to First Deterioration (CAT, SGRQ, TDI, EXAC (mod/sev)) (Days) | | SAC |
| Rescue ( | Use | | | |
| 2.65 | ITT | Least Squares Mean (95% CI) Change from Baseline in Percentage of Rescue-Free Days over Weeks 1-24 using e-Diary | | SAC |
| 2.66 | ITT | Least Squares Mean (95% CI) Change from Baseline in Percentage of Rescue-Free Days over Weeks 1-24 using eMDI | | SAC |
| Physical | Activity Mo | onitor | | |
| 2.67 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Step Count | | SAC |
| 2.68 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Duration of Light Physical Activity Duration(Hours) | | SAC |

| Efficacy: | Efficacy: Figures | | | |
|---|---|---|---|---|
| | Popu-<br>lation | Title | Programming Note | Deliverable |
| 2.69 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Duration of Moderate to Vigorous Physical Activity (Hours) | | SAC |
| 2.70 | ITT | Least Squares Mean (95% CI) Change from Baseline in Weekly Mean Total Energy Expenditure (kCal) | | SAC |

# 10.8.4. Safety Tables

| Safety Tables | | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| Exposure | • | • | | |
| 3.34 | ITT | Summary of Exposure | | SAC |
| Adverse Ev | ents | | | |
| 3.35 | ITT | Overview of Adverse Events | | SAC |
| 3.36 | ITT | Summary of On-treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.37 | ITT | Summary of On-treatment Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.38 | ITT | Summary of On-treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |

| Safety Tables | | | | |
|---|---|---|---|---|
| No. | Popu-<br>lation | Title | Programming Note | Deliverable |
| 3.39 | ITT | Summary of On-treatment Fatal Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.40 | ITT | Summary of Common (>=3%) On-treatment Non-serious Drug-related Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 3.41 | ITT | Summary of Common (>=3%) On-treatment Serious Adverse Events by Overall Frequency | | SAC |
| 3.42 | ITT | Summary of Common (>=3%) On-treatment Serious Drug-related Adverse Events by Overall Frequency | | SAC |